CLINICAL TRIAL: NCT03544281
Title: A Phase I/II, Open-label, Dose Escalation and Expansion Study to Evaluate Safety, Tolerability, and Clinical Activity of the Antibody-Drug Conjugate GSK2857916 Administered in Combination With Lenalidomide Plus Dexamethasone (Arm A), or Bortezomib Plus Dexamethasone (Arm B) in Participants With Relapsed / Refractory Multiple Myeloma - DREAMM-6
Brief Title: To Evaluate Safety, Tolerability, and Clinical Activity of the Antibody-drug Conjugate, GSK2857916 Administered in Combination With Lenalidomide Plus Dexamethasone (Arm A), or in Combination With Bortezomib Plus Dexamethasone (Arm B) in Participants With Relapsed/Refractory Multiple Myeloma (RRMM)
Acronym: DREAMM 6
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 207497; 2017-004689-93 (EudraCT Number)
Record Dates: First submitted 2018-04-30; First posted 2018-06-01 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
Keywords: Relapsed / Refractory Multiple Myeloma; Antibody-Drug Conjugate; belantamab mafodotin; Combination therapy; Belamaf
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; Lenalidomide; Dexamethasone; Bortezomib

STUDY DESIGN:
Masking Description: This is an open-label study; therefore, no blinding of treatment identity will be done for both treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Belantamab mafodotin+lenalidomide +dexamethasone (Experimental): Participants will receive SINGLE full dose of belantamab mafodotin as 2.5 mg/kg and 1.9 mg/kg on Day 1 of every 28-day cycle as a 30-60 min infusion.
  SPLIT: belantamab mafodotin will be administered in two equal divided doses, 2.5 mg/kg SPLIT dose of a 1.25 mg/kg dose on Day 1 and a 1.25 mg/kg dose on Day 8 of each 28-day cycle.
  STRETCH: belantamab mafodotin will be administered as 1.9 mg/kg dose on Day 1 of every alternate 28-day cycles (C1, C3, C5, C7 and so on.) Participants will also receive Lenalidomide 25 mg or 10 mg orally daily, on Days 1-21 of each 28 day cycle with Dexamethasone, 40 mg weekly per oral (PO)/intravenously (IV) on Days 1,8,15, & 22 of each cycle.
  Interventions: Drug: Belantamab mafodotin; Drug: Lenalidomide; Drug: Dexamethasone
- Arm B: Belantamab mafodotin+bortezomib+dexamethasone (Experimental): Participants will receive SINGLE full dose of belantamab mafodotin as 3.4 mg/kg; 2.5 mg/kg; 1.9 mg/kg on Day 1 of each 21-day cycle. SPLIT: belantamab mafodotin will be administered in two equal divided doses: 3.4 mg/kg SPLIT as 1.7 mg/kg dose on Day 1 & 1.7 mg/kg dose on Day 8; 2.5 mg/kg SPLIT dosing as 1.25 mg/kg dose on Day 1 & 1.25 mg/kg dose on Day 8 of each 21-day cycle. STRETCH: belantamab mafodotin will be administered as single dose of 2.5 mg/kg on Day 1 of every alternate 21-day cycles (C1,C3,C5,C7 & so on), 1.9 mg/kg administered on Day 1 of every alternate 21-day cycles (C1,C3,C5,C7 and so on). Step Down(S/D) STRETCH=belantamab mafodotin 2.5 mg/kg dose will be administered on Day 1 C1 followed by 1.9 mg/kg starting dose on Day1 of alternate 21-day cycles C3 onwards (C3,C5,C7, & so on). Bortezomib will be administered at 1.3 mg/m^2 SC/IV on Days 1,4,8, & 11 of every 21-day cycle. Dex will be administered at 20 mg PO or IV on Days 1,2,4,5,8,9,11, & 12 of every 21-day cycle.
  Interventions: Drug: Belantamab mafodotin; Drug: Dexamethasone; Drug: Bortezomib

INTERVENTIONS:
Drug: Belantamab mafodotin — Selected doses of belantamab mafodotin will be administered as an infusion.
Drug: Lenalidomide — Lenalidomide will be administered as 25 or 10 mg,orally, with belantamab mafodotin and dexamethasone.
  Arms: Arm A: Belantamab mafodotin+lenalidomide +dexamethasone
Drug: Dexamethasone — Dexamethasone will be administered as 20 or 40 mg, orally with belantamab mafodotin.
Drug: Bortezomib — Bortezomib will be administered as 1.3 mg/m^2, as SC or IV, with belantamab mafodotin and dexamethasone.
  Arms: Arm B: Belantamab mafodotin+bortezomib+dexamethasone

SUMMARY:
This study will evaluate the safety and tolerability profile of belantamab mafodotin when administered in combination with approved regimens of either Lenalidomide Plus Dexamethasone [Len/Dex (Treatment A)] or Bortezomib Plus Dexamethasone [Bor/Dex (Treatment B)] in participants with RRMM, i.e., those who have relapsed or who are refractory to at least 1 line of approved therapy.

Participants receiving treatment A, may continue combination treatment until the occurrence of progressive disease (PD), intolerable adverse events (AEs ), consent withdrawal, death or end of study. The participants receiving treatment B, may continue combination treatment for a total of up to 8 cycles. After 8 cycles of combination therapy, the participants will continue treatment with belantamab mafodotin, as a monotherapy until the occurrence of PD, intolerable AEs, consent withdrawal, death or end of study.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent.
* Male or female, 18 years or older (at the time consent is obtained).
* Have confirmed diagnosis of Multiple Myeloma (MM) as defined by the IMWG.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 for Arm A and 0 to 2 for Arm B.
* Have undergone stem cell transplant (SCT), or are considered transplant ineligible.
* Have been previously treated with at least 1 prior line of MM therapy, and must have documented disease progression during or after their most recent therapy.
* Must have at least ONE aspect of measurable disease, defined as one the following: Urine M-protein excretion >=200 milligram (mg)/24 hours, or; Serum M-protein concentration >=0.5 gram (g)/deciliter (dL) (>=5.0 g/Liter), or; Serum free light chain (FLC) assay: involved FLC level >=10 mg/dL (>=100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65).
* Participants with a history of autologous SCT, are eligible for study participation provided the following eligibility criteria are met: Autologous SCT was >100 days prior to study enrollment; No active bacterial, viral, or fungal infection(s) present; Participant meets the remainder of the eligibility criteria.
* All prior treatment-related toxicities (defined by National Cancer Institute Common Toxicity Criteria for Adverse Events [NCI-CTCAE], Version 4.03, 2010) must be Grade <= 1 at the time of enrollment, except for alopecia. Participants with Grade 2 neuropathy can be enrolled into Len/Dex treatment arm, but not into Bor/Dex treatment arm.
* Adequate organ system functions as defined by the laboratory assessments.
* The contraceptions used by female participants be consistent with local regulations, regarding methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: is not a woman of child bearing potential (WOCBP) or Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency, during the intervention period and for at least 4 months after the last dose of belantamab mafodotin and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

WOCBP Participants Assigned to Arm A:

* Due to lenalidomide being a thalidomide analogue with risk for embryo-fetal toxicity and prescribed under a pregnancy prevention/controlled distribution program, WOCBP participants will be eligible if they commit either to abstain continuously from heterosexual sexual intercourse or to use two methods of reliable birth control (one method that is highly effective; beginning 4 weeks prior to initiating treatment with lenalidomide, during therapy, during dose interruptions and continuing for 4 weeks following discontinuation of lenalidomide treatment. Thereafter, WOCBP participants must use a contraceptive method that is highly effective (with a failure rate of <1% per year) for a further 3 months, and agree not to donate eggs (ova, oocytes) for the purpose of reproduction during this period: Two negative pregnancy tests must be obtained prior to initiating lenalidomide therapy. The first test should be performed within 10-14 days and the second test within 24 hours prior to prescribing lenalidomide therapy.

WOCBP Participants Assigned to Arm B

* WOCBP assigned to Arm B must have a negative highly sensitive serum pregnancy test within 72 hours of dosing on C1D1 and agree to use effective contraception during the study and for 4 months after the last dose of belantamab mafodotin or 7 months from the last dose of bortezomib, whichever is longer.
* Male participants using contraception should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Male participants are eligible to participate if they agree to the following:

Arm A: from the time of first dose of study until 6 months after the last dose of belantamab mafodotin 4 weeks after the last dose of lenalidomide, whichever is longer, to allow for clearance of any altered sperm.

Arm B: from the time of first dose of study until 6 months after the last dose of belantamab mafodotin or 4 months from the last dose of bortezomib (whichever is the longer) to allow for clearance of any altered sperm.

* Male participants must agree to refrain from donating sperm and either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR Must agree to use contraception/barrier as detailed below.
* Agree to use a male condom even if they have undergone a successful vasectomy and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year when having sexual intercourse. Male participants should also use a condom with pregnant females. If the female partner of the male participant is pregnant at the time of enrollment, or becomes pregnant during the trial, the male participant must agree to remain abstinent (if it is consistent with their preferred and usual lifestyle) or use a male condom.

Exclusion Criteria:

* Systemic anti-myeloma therapy (including systemic steroids) within <=14 days, or plasmapheresis within 7 days prior to the first dose of study drug.
* Use of an investigational drug within 14 days or five half-lives (whichever is longer) preceding the first dose of study drug.
* Prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drugs.
* Prior allogenic stem cell transplant. Note: Participants who have undergone syngeneic transplant will be allowed only if they have no history and no currently active, graft versus host disease (GvHD).
* Evidence of active mucosal or internal bleeding.
* Any major surgery within the last four weeks.
* Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM are eligible, provided they fulfill criteria.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, or otherwise stable chronic liver disease per investigator's assessment).
* Participants with invasive malignancies other than multiple myeloma are excluded, unless the second malignancy has been considered medically stable for at least 2 years. The participant must not be receiving active therapy, other than hormonal therapy for this disease. Note: Participants with curatively treated non-melanoma skin cancer are allowed without a 2-year restriction.
* Evidence of cardiovascular risk including any of the following: Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities including 2nd degree (Type II) or 3rd degree atrioventricular (AV) block; History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months of Screening; Class III or IV heart failure as defined by the New York Heart Association functional classification system; Uncontrolled hypertension.
* Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
* Pregnant or lactating female.
* Active infection requiring treatment.
* Known Human immunodeficiency virus (HIV) infection.
* Presence of hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb at Screening or within 3 months prior to first dose of study treatment).
* Current corneal disease except for mild punctuate keratopathy.
* Positive hepatitis C antibody test result or positive hepatitis C Ribonucleic acid (RNA) test result at Screening or within 3 months prior to first dose of study treatment.
* Current corneal disease except for mild punctute keratopathy.
* Participants Assigned to Treatment A (belantamab mafodotin plus Len/Dex): Participants unable to tolerate antithrombotic prophylaxis must be excluded; Discontinuation of prior treatment with lenalidomide due to intolerable AEs.
* Participants Assigned to Treatment B (belantamab mafodotin plus Bor/Dex): Unacceptable AEs from previous bortezomib treatment; Ongoing Grade 2 or higher peripheral neuropathy or neuropathic pain from previous bortezomib treatment; Intolerance or contraindications to anti-viral prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- United States (12):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Goodyear, Arizona
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Grand Island, Nebraska
  - GSK Investigational Site, Hackensack, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Dallas, Texas
- Australia (6):
  - GSK Investigational Site, Wollongong, New South Wales
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Murdoch, Western Australia
  - GSK Investigational Site, Nedlands, Western Australia
- GSK Investigational Site, Montreal, Quebec, Canada
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Salamanca
- United Kingdom (2):
  - GSK Investigational Site, Truro, Cornwall
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of two phases - Main Study Phase (Day 1 to Month 53) and Post Analysis Continued Treatment (PACT) Phase (From Month 53 up to Month 65, which marks the completion of the PACT Phase for all participants). In PACT phase those participants still benefiting from drug continued to receive study drug until discontinued or withdrawn from study.
Groups:
- Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex: Participants with Relapsed or Refractory Multiple Myeloma (RRMM) received belantamab mafodotin as 1.9 milligram (mg)/kilogram (kg) dose on Day 1 of every alternate 28-day cycles (C1, C3, C5, C7 and so on) as a 30-60 minute infusion. Along with belantamab mafodotin, Lenalidomide (Len) was administered as 25 mg or 10 mg per oral (PO) on Days 1-21 of each 28-day cycle with 40 mg Dexamethasone (Dex) weekly PO/ intravenously (IV) on Days 1, 8, 15 and 22 of each cycle.
- Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex: Participants with RRMM received belantamab mafodotin as SINGLE full dose of 1.9 mg/kg on Day 1 of every 28-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Lenalidomide was administered as 25 mg or 10 mg PO on Days 1-21 of each 28-day cycle with 40 mg Dexamethasone weekly PO/ IV on Days 1, 8, 15 and 22 of each cycle.
- Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex: Participants with RRMM received belantamab mafodotin as two equal divided doses of a total 2.5mg/kg dose as a 1.25 mg/kg dose on Day 1 and a 1.25 mg/kg dose on Day 8 of each 28-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Lenalidomide was administered as 25 mg or 10 mg PO on Days 1-21 of each 28-day cycle with 40 mg Dexamethasone weekly PO/ IV on Days 1, 8, 15 and 22 of each cycle.
- Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex: Participants with RRMM received belantamab mafodotin as SINGLE full dose of 2.5 mg/kg on Day 1 of every 28-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Lenalidomide was administered as 25 mg or 10 mg PO on Days 1-21 of each 28-day cycle with 40 mg Dexamethasone weekly PO/ IV on Days 1, 8, 15 and 22 of each cycle.
- Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex: Participants with RRMM received belantamab mafodotin as 1.9 mg/kg dose on Day 1 of every alternate 21-day cycle (C1, C3, C5, C7, and so on) as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib (Bor) was administered as 1.3 milligrams per square meters (mg/m^2) subcutaneously (SC) /IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone (Dex) PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles.
- Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex: Participants with RRMM received belantamab mafodotin as SINGLE full dose of 1.9 mg/kg on Day 1 of every 21-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC /IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles.
- Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex: Participants with RRMM received belantamab mafodotin as 2.5 mg/kg dose on cycle 1 day 1 (C1D1) followed by 1.9 mg/kg step-down dose on Day 1 of every alternate 21-day cycles C3 onwards (C3, C5, C7, and so on) as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC /IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles.
- Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex: Participants with RRMM received belantamab mafodotin as 2.5 mg/kg dose on Day 1 of every alternate 21-day cycles (C1, C3, C5, C7, and so on) as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC /IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles.
- Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex: Participants with RRMM received belantamab mafodotin as two equal divided doses of a total 2.5mg/kg dose as a 1.25 mg/kg on Day 1 and 1.25 mg/kg dose on Day 8 of every 21-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC /IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles.
- Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex: Participants with RRMM received belantamab mafodotin as SINGLE full dose of 2.5 mg/kg on Day 1 of every 21-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC /IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles.
- Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex: Participants with RRMM received belantamab mafodotin as two equal divided doses of a total 3.4 mg/kg dose as a 1.7 mg/kg dose on Day 1 and 1.7 mg/kg on Day 8 of every 21-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC /IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles.
- Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex: Participants with RRMM received belantamab mafodotin as SINGLE full dose of 3.4 mg/kg on Day 1 of every 21-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC /IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles.
- PACT Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex: Participants with Relapsed or Refractory Multiple Myeloma (RRMM) received belantamab mafodotin as 1.9 milligram (mg)/kilogram (kg) dose on Day 1 of every alternate 28-day cycles (C1, C3, C5, C7 and so on) as a 30-60 minute infusion. Along with belantamab mafodotin, Lenalidomide (Len) was administered as 25 mg or 10 mg per oral (PO) on Days 1-21 of each 28-day cycle with 40 mg Dexamethasone (Dex) weekly PO/ intravenously (IV) on Days 1, 8, 15 and 22 of each cycle until PD, death, intolerable toxicity, or consent withdrawn.
- PACT Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex: Participants with RRMM received belantamab mafodotin as SINGLE full dose of 1.9 mg/kg on Day 1 of every 28-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Lenalidomide was administered as 25 mg or 10 mg PO on Days 1-21 of each 28-day cycle with 40 mg Dexamethasone weekly PO/ IV on Days 1, 8, 15 and 22 of each cycle until PD, death, intolerable toxicity, or consent withdrawn.
- PACT Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex: Participants with RRMM received belantamab mafodotin as two equal divided doses of a total 2.5mg/kg dose as a 1.25 mg/kg dose on Day 1 and a 1.25 mg/kg dose on Day 8 of each 28-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Lenalidomide was administered as 25 mg or 10 mg PO on Days 1-21 of each 28-day cycle with 40 mg Dexamethasone weekly PO/ IV on Days 1, 8, 15 and 22 of each cycle until PD, death, intolerable toxicity, or consent withdrawn.
- PACT Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex: Participants with RRMM received belantamab mafodotin as SINGLE full dose of 2.5 mg/kg on Day 1 of every 28-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Lenalidomide was administered as 25 mg or 10 mg PO on Days 1-21 of each 28-day cycle with 40 mg Dexamethasone weekly PO/ IV on Days 1, 8, 15 and 22 of each cycle until PD, death, intolerable toxicity, or consent withdrawn.
- PACT Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex: Participants with RRMM received belantamab mafodotin as 1.9 mg/kg dose on Day 1 of every alternate 21-day cycle (C1, C3, C5, C7, and so on) as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib (Bor) was administered as 1.3 milligrams per square meters (mg/m^2) subcutaneously (SC) /IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone (Dex) PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles followed by belantamab mafodotin monotherapy as 1.9 mg/kg dose until PD, death, intolerable toxicity, or consent withdrawn.
- PACT Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex: Participants with RRMM received belantamab mafodotin as SINGLE full dose of 1.9 mg/kg on Day 1 of every 21-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC /IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles followed by belantamab mafodotin monotherapy as 1.9 mg/kg dose until PD, death, intolerable toxicity, or consent withdrawn.
- PACT Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex: Participants with RRMM received belantamab mafodotin as 2.5 mg/kg dose on cycle 1 day 1 (C1D1) followed by 1.9 mg/kg step-down dose on Day 1 of every alternate 21-day cycles C3 onwards (C3, C5, C7, and so on) as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC /IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles followed by belantamab mafodotin monotherapy as 2.5 mg/kg dose until PD, death, intolerable toxicity, or consent withdrawn.
- PACT Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex: Participants with RRMM received belantamab mafodotin as two equal divided doses of a total 2.5mg/kg dose as a 1.25 mg/kg on Day 1 and 1.25 mg/kg dose on Day 8 of every 21-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC /IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles followed by belantamab mafodotin monotherapy as 2.5 mg/kg dose until PD, death, intolerable toxicity, or consent withdrawn.
- PACT Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex: Participants with RRMM received belantamab mafodotin as SINGLE full dose of 2.5 mg/kg on Day 1 of every 21-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC /IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles followed by belantamab mafodotin monotherapy as 2.5 mg/kg dose until PD, death, intolerable toxicity, or consent withdrawn.
- PACT Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex: Participants with RRMM received belantamab mafodotin as two equal divided doses of a total 3.4 mg/kg dose as a 1.7 mg/kg dose on Day 1 and 1.7 mg/kg on Day 8 of every 21-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC /IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles followed by belantamab mafodotin monotherapy as 3.4 mg/kg dose until PD, death, intolerable toxicity, or consent withdrawn.
Period: Main Study Phase
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex | PACT Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | PACT Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | PACT Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | PACT Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | PACT Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | PACT Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | PACT Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | PACT Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | PACT Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | PACT Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex
Started | 12 | 4 | 13 | 16 | 12 | 12 | 13 | 12 | 13 | 18 | 12 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
All Treated (All participants who received at least one dose of study treatment.) | 12 | 4 | 13 | 16 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DLT-evaluable (DLT-evaluable population included participants who received at least 1 full dose of belantamab mafodotin and at least 75% of planned doses of Len/Dex by the end of Cycle 1 (Day 28) for treatment A and participants who received at least 1 full dose of belantamab mafodotin and at least 75% of planned doses of Bor/Dex by the end of Cycle 1 (Day 21) for treatment B.) | 0 | 3 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Participants who completed main study.) | 4 | 1 | 4 | 2 | 6 | 6 | 4 | 6 | 4 | 4 | 4 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 3 | 9 | 14 | 6 | 6 | 9 | 6 | 9 | 14 | 8 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 3 | 2 | 6 | 8 | 4 | 2 | 4 | 5 | 5 | 8 | 6 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Ongoing | 3 | 1 | 2 | 4 | 2 | 4 | 4 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator Site Closed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did not receive study treatment | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PACT Phase
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex | PACT Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | PACT Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | PACT Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | PACT Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | PACT Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | PACT Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | PACT Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | PACT Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | PACT Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | PACT Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 4 | 2 | 4 | 4 | 2 | 2 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 4 | 2 | 3 | 3 | 2 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated population included all participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex | Total
Number analyzed (Participants) | 12 | 4 | 13 | 16 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16 | 152
Age, Customized [Count of Participants; unit: Participants]
  18 to <65 years | 4 | 3 | 4 | 4 | 6 | 3 | 4 | 4 | 5 | 6 | 6 | 9 | 58
  65 to <75 years | 5 | 1 | 8 | 8 | 3 | 8 | 7 | 4 | 5 | 8 | 5 | 5 | 67
  >=75 years | 3 | 0 | 1 | 4 | 3 | 1 | 1 | 4 | 3 | 4 | 1 | 2 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 5 | 3 | 5 | 3 | 5 | 7 | 2 | 7 | 4 | 5 | 48
  Male | 10 | 4 | 8 | 13 | 7 | 9 | 7 | 5 | 11 | 11 | 8 | 11 | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 4 | 0 | 1 | 10
  Asian - Central/South Asian Heritage | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Asian - East Asian Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian - South East Asian Heritage | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  White - Arabic/North African Heritage | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  White - White/Caucasian/European Heritage | 11 | 4 | 13 | 13 | 11 | 11 | 10 | 7 | 11 | 12 | 11 | 15 | 129
  Missing | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs), Treatment A
Description: DLT is an adverse event (AE) that is considered by the investigator to be clinically relevant and attributed to the study therapy during the 28 day DLT period and meets at least one of the DLT criteria: Grade 3 or greater febrile neutropenia lasting >48 hours (h) despite adequate treatment; Grade 4 thrombocytopenia <25,000/mm^3 accompanied by significant bleeding; any Grade 3 or greater non-hematologic laboratory value (if laboratory abnormality persist >48 h despite supportive treatment or abnormality leading to hospitalisation); non-hematologic toxicity which does not resolve with appropriate supportive treatment within 48 h, Grade 4 corneal adverse events; and other organ specific toxicities (liver toxicity that causes discontinuation of treatment).
Time Frame: Up to 28 days
Population: DLT-evaluable population included participants who received at least 1 full dose of belantamab mafodotin and at least 75% of planned doses of Len/Dex by the end of Cycle 1 (Day 28). As pre-specified in protocol, only specified treatment arms were planned to be analyzed for DLTs.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 3 | 4 | 6
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants With DLTs, Treatment B
Description: DLT is an adverse event (AE) that is considered by the investigator to be clinically relevant and attributed to the study therapy during the 21 day DLT period and meets at least one of the DLT criteria: Grade 3 or greater febrile neutropenia lasting >48 hours (h) despite adequate treatment; Grade 4 thrombocytopenia <25,000/mm^3 accompanied by significant bleeding; any Grade 3 or greater non-hematologic laboratory value (if laboratory abnormality persist >48 h despite supportive treatment or abnormality leading to hospitalisation); non-hematologic toxicity which does not resolve with appropriate supportive treatment within 48 h, Grade 4 corneal adverse events; and other organ specific toxicities (liver toxicity that causes discontinuation of treatment).
Time Frame: Up to 21 days
Population: DLT-evaluable population included participants who received at least 1 full dose of belantamab mafodotin and at least 75% of planned doses of Bor/Dex by the end of Cycle 1 (Day 21). As pre-specified in protocol, only specified treatment arms were planned to be analyzed for DLTs.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 6 | 7
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose results in death, Is life-threatening, Requires inpatient hospitalization or prolongation of existing hospitalization, Results in persistent disability/incapacity or Is a congenital anomaly/birth defect, Other situations which involve medical or scientific judgment or is associated with liver injury and impaired liver function. SAEs are subset of AEs. A summary of number of participants with any AEs and SAEs are presented. AEs were coded using the Medical Dictionary for Regulatory Affairs (MedDRA dictionary).
Time Frame: Up to approximately 4.5 years
Population: All treated population included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Participants
  Any AE | 12 | 4 | 13 | 16 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Any SAE | 6 | 2 | 6 | 10 | 8 | 8 | 6 | 6 | 7 | 13 | 6 | 9

4. Primary Outcome: Number of Participants With Worst-Case Amount of Increase From Baseline Value in Corrected QT Interval Using Fredericia's Formula (QTcF)
Description: 12-lead electrocardiogram (ECGs) were obtained using an automated ECG machine that automatically calculated the QTcF intervals. QTc values are categorized into the clinical concern ranges which are specific to changes in QTc: 31-60 milliseconds (msec), and >60 msec, and >530msec. An increase is defined relative to Baseline. Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits. Data of number of participants with worst-case increase post baseline is presented.
Time Frame: Up to approximately 4.5 years
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16 | 10 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Participants
  Increase of 31-60 msec | 3 | 3 | 5 | 3 | 1 | 3 | 1 | 2 | 5 | 4 | 5 | 5
  Increase of >60 msec | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  Increase of >530 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Worst-case Grade Change From Baseline in Hematology Parameters
Description: Blood samples were collected for analysis of following hematology parameters: Hemoglobin (hemoglobin increased and anemia), Lymphocytes (lymphocyte count increased and lymphocyte count decreased), Neutrophils, Platelets and Leukocytes (leukocytosis and white blood cells decreased). The laboratory parameters were graded according to Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.03. Grade (G) 1: mild; G2: moderate; G3: severe or medically significant; G4: life-threatening consequences. Higher grade indicates greater severity and increase in grade was defined relative to Baseline grade. Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits. Any worst-case post baseline increases in grade along with any increase to a maximum G3 and a maximum G4 are presented.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Participants
  Hemoglobin increased, Any Grade Increase | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  Hemoglobin increased, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia, Any Grade Increase | 7 | 2 | 8 | 9 | 5 | 6 | 2 | 3 | 9 | 11 | 8 | 10
  Anemia, Increase to Grade 3 | 0 | 0 | 3 | 2 | 2 | 2 | 1 | 2 | 5 | 2 | 2 | 3
  Anemia, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Lymphocyte count increased, Any Grade Increase | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocyte count increased, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Lymphocyte count increased, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Lymphocyte count increased, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Lymphocyte count decreased, Any Grade Increase | 11 | 3 | 10 | 12 | 11 | 12 | 10 | 11 | 12 | 13 | 10 | 15
  Lymphocyte count decreased, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Lymphocyte count decreased, Increase to Grade 3 | 7 | 1 | 3 | 4 | 5 | 6 | 3 | 5 | 6 | 6 | 3 | 8
  Lymphocyte count decreased, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Lymphocyte count decreased, Increase to Grade 4 | 0 | 0 | 1 | 3 | 1 | 3 | 2 | 1 | 3 | 2 | 3 | 1
  Neutrophils, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 15 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Neutrophils, Any Grade Increase | 8 | 3 | 9 | 9 | 6 | 6 | 5 | 4 | 7 | 10 | 8 | 9
  Neutrophils, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 15 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Neutrophils, Increase to Grade 3 | 3 | 2 | 4 | 4 | 1 | 3 | 3 | 1 | 3 | 1 | 4 | 2
  Neutrophils, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 15 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Neutrophils, Increase to Grade 4 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0
  Platelets, Any Grade Increase | 9 | 4 | 12 | 15 | 11 | 12 | 11 | 12 | 13 | 18 | 12 | 16
  Platelets, Increase to Grade 3 | 1 | 1 | 4 | 5 | 3 | 2 | 4 | 3 | 5 | 3 | 2 | 3
  Platelets, Increase to Grade 4 | 1 | 0 | 2 | 1 | 7 | 9 | 5 | 6 | 6 | 9 | 9 | 10
  Leukocytosis, Any Grade Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased, Any Grade Increase | 10 | 3 | 11 | 8 | 5 | 8 | 3 | 7 | 8 | 11 | 8 | 13
  White blood cell decreased, Increase to Grade 3 | 2 | 0 | 1 | 3 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 0
  White blood cell decreased, Increase to Grade 4 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Worst-case Change Post-baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of following hematology parameters: basophils, eosinophils, hematocrit, mean corpuscular hemoglobin concentration (MCHC), mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), monocytes, erythrocytes and reticulocyte. The summaries of worst-case change from baseline with respect to normal range was analyzed for only those laboratory tests that were not gradable by CTCAE version 4.03. The number of participants with decreases to low from baseline, changes to normal or no changes from baseline, and increases to high values from baseline have been presented. Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All treated population. Only those participants with data available at specified time points have been analyzed. Participants are counted twice if the participant has values that changed "Decreased to Low" and "Increased to High", so the sum of the percentages may not add to 100% for each category.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Participants
  Basophils, Decrease to Low: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Basophils, Decrease to Low | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Basophils, Change to Normal or No Change: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Basophils, Change to Normal or No Change | 10 | 4 | 10 | 10 | 9 | 10 | 10 | 11 | 11 | 12 | 11 | 12
  Basophils, Increase to High: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Basophils, Increase to High | 2 | 0 | 3 | 4 | 2 | 1 | 2 | 1 | 2 | 2 | 1 | 1
  Eosinophils, Decrease to Low: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Eosinophils, Decrease to Low | 2 | 1 | 4 | 2 | 1 | 3 | 0 | 2 | 3 | 2 | 1 | 2
  Eosinophils, Change to Normal or No Change: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Eosinophils, Change to Normal or No Change | 7 | 2 | 8 | 7 | 11 | 9 | 12 | 10 | 10 | 11 | 10 | 13
  Eosinophils, Increase to High: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Eosinophils, Increase to High | 3 | 2 | 3 | 6 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0
  Hematocrit, Decrease to Low | 4 | 1 | 1 | 4 | 2 | 5 | 1 | 1 | 3 | 3 | 1 | 7
  Hematocrit, Change to Normal or No Change | 8 | 3 | 12 | 12 | 10 | 7 | 9 | 11 | 10 | 14 | 11 | 8
  Hematocrit, Increase to High | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1
  MCH, Decrease to Low | 0 | 0 | 3 | 1 | 0 | 3 | 1 | 3 | 2 | 6 | 2 | 1
  MCH, Change to Normal or No Change | 9 | 3 | 7 | 13 | 10 | 7 | 8 | 9 | 10 | 9 | 10 | 11
  MCH, Increase to High | 3 | 1 | 3 | 2 | 2 | 3 | 3 | 0 | 1 | 4 | 0 | 4
  MCHC, Decrease to Low | 4 | 0 | 4 | 4 | 2 | 6 | 5 | 6 | 6 | 7 | 5 | 5
  MCHC, Change to Normal or No Change | 8 | 3 | 9 | 12 | 8 | 6 | 6 | 6 | 6 | 10 | 6 | 11
  MCHC, Increase to High | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 2 | 1 | 0
  MCV, Decrease to Low | 0 | 0 | 4 | 1 | 0 | 2 | 1 | 2 | 0 | 4 | 0 | 0
  MCV, Change to Normal or No Change | 10 | 3 | 7 | 11 | 10 | 7 | 7 | 10 | 11 | 10 | 10 | 13
  MCV, Increase to High | 2 | 1 | 3 | 4 | 2 | 3 | 5 | 1 | 2 | 4 | 2 | 3
  Monocytes, Decrease to Low: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Monocytes, Decrease to Low | 5 | 1 | 4 | 3 | 5 | 4 | 7 | 8 | 5 | 7 | 3 | 5
  Monocytes, Change to Normal or No Change: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Monocytes, Change to Normal or No Change | 4 | 2 | 2 | 4 | 3 | 1 | 1 | 1 | 2 | 3 | 5 | 4
  Monocytes, Increase to High: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 15 | 12 | 15
  Monocytes, Increase to High | 4 | 2 | 11 | 10 | 6 | 10 | 10 | 8 | 8 | 10 | 5 | 8
  Erythrocytes, Decrease to Low | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 4 | 2 | 3
  Erythrocytes, Change to Normal or No Change | 9 | 3 | 13 | 13 | 11 | 10 | 12 | 11 | 13 | 14 | 9 | 13
  Erythrocytes, Increase to High | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
  Reticulocytes, Decrease to Low: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Reticulocytes, Decrease to Low | 3 | 1 | 2 | 4 | 1 | 1 | 2 | 4 | 2 | 4 | 3 | 5
  Reticulocytes, Change to Normal or No Change: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Reticulocytes, Change to Normal or No Change | 7 | 1 | 5 | 7 | 9 | 6 | 5 | 2 | 8 | 6 | 4 | 2
  Reticulocytes, Increase to High: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Reticulocytes, Increase to High | 3 | 2 | 7 | 6 | 2 | 6 | 7 | 8 | 3 | 9 | 6 | 10

7. Primary Outcome: Number of Participants With Worst-case Grade Change From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for analysis of following clinical chemistry parameters: Hyperglycemia, Hypoglycemia, Albumin, Alkaline Phosphatase, Alanine Aminotransferase (ALT), Aspartate Aminotransferase, (AST), Bilirubin, Creatine Kinase (CK), Creatinine, Gamma Glutamyl Transferase (GGT), Hyperkalemia, Hypokalemia, Hypermagnesemia, Hypomagnesemia, Phosphate, Hypernatremia, Hyponatremia, Urate, Hypercalcemia and Hypocalcemia. Laboratory parameters were graded according to CTCAE v4.03. Grade (G) 1: mild; G2: moderate; G3: severe or medically significant; G4: life-threatening consequences. Higher grade indicates greater severity and increase in grade was defined relative to Baseline grade. Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits. Any worst-case post baseline increases in grade along with any increase to a maximum G3 and a maximum G4 are presented.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 15 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Participants
  Hyperglycemia, Any Grade Increase: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 12 | 18 | 12 | 16
  Hyperglycemia, Any Grade Increase | 3 | 1 | 9 | 11 | 8 | 9 | 9 | 8 | 5 | 10 | 6 | 8
  Hyperglycemia, Increase to Grade 3: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 12 | 18 | 12 | 16
  Hyperglycemia, Increase to Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 1
  Hyperglycemia, Increase to Grade 4: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 12 | 18 | 12 | 16
  Hyperglycemia, Increase to Grade 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Hypoglycemia, Any Grade Increase: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 12 | 18 | 12 | 16
  Hypoglycemia, Any Grade Increase | 2 | 0 | 1 | 1 | 0 | 2 | 1 | 3 | 0 | 1 | 0 | 1
  Hypoglycemia, Increase to Grade 3: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 12 | 18 | 12 | 16
  Hypoglycemia, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypoglycemia, Increase to Grade 4: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 12 | 18 | 12 | 16
  Hypoglycemia, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin, Any Grade Increase | 6 | 2 | 8 | 9 | 5 | 8 | 4 | 5 | 7 | 14 | 5 | 8
  Albumin, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 0
  Albumin, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Alkaline Phosphatase, Any Grade Increase | 4 | 0 | 7 | 6 | 6 | 4 | 5 | 6 | 8 | 8 | 2 | 5
  Alkaline Phosphatase, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Alkaline Phosphatase, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Alkaline Phosphatase, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  ALT, Any Grade Increase | 7 | 1 | 7 | 7 | 5 | 5 | 9 | 8 | 6 | 6 | 7 | 8
  ALT, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  ALT, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1
  ALT, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  ALT, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  AST, Any Grade Increase: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  AST, Any Grade Increase | 4 | 2 | 8 | 6 | 10 | 12 | 8 | 10 | 8 | 11 | 8 | 12
  AST, Increase to Grade 3: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  AST, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0
  AST, Increase to Grade 4: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  AST, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Bilirubin, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Bilirubin, Any Grade Increase | 1 | 0 | 1 | 4 | 2 | 2 | 0 | 3 | 2 | 2 | 1 | 5
  Bilirubin, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Bilirubin, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Bilirubin, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CK, Any Grade Increase: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  CK, Any Grade Increase | 3 | 2 | 4 | 2 | 1 | 3 | 3 | 4 | 4 | 4 | 4 | 7
  CK, Increase to Grade 3: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  CK, Increase to Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  CK, Increase to Grade 4: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  CK, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Creatinine, Any Grade Increase | 1 | 0 | 7 | 2 | 2 | 2 | 6 | 2 | 4 | 3 | 1 | 6
  Creatinine, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Creatinine, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Creatinine, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GGT, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  GGT, Any Grade Increase | 9 | 1 | 9 | 9 | 6 | 7 | 5 | 10 | 8 | 10 | 6 | 9
  GGT, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  GGT, Increase to Grade 3 | 2 | 0 | 2 | 4 | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 2
  GGT, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  GGT, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hyperkalemia, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hyperkalemia, Any Grade Increase | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 3 | 3 | 0 | 3
  Hyperkalemia, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hyperkalemia, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hyperkalemia, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hypokalemia, Any Grade Increase | 3 | 2 | 3 | 4 | 6 | 4 | 8 | 3 | 4 | 6 | 7 | 4
  Hypokalemia, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hypokalemia, Increase to Grade 3 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Hypokalemia, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hypokalemia, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hypermagnesemia, Any Grade Increase | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 4 | 1 | 1 | 2
  Hypermagnesemia, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hypermagnesemia, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Hypermagnesemia, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hypermagnesemia, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hypomagnesemia, Any Grade Increase | 3 | 2 | 3 | 4 | 3 | 2 | 0 | 1 | 1 | 7 | 4 | 4
  Hypomagnesemia, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hypomagnesemia, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hypomagnesemia, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Phosphate, Any Grade Increase: number analyzed (Participants) | 11 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Phosphate, Any Grade Increase | 6 | 3 | 5 | 4 | 4 | 7 | 6 | 5 | 8 | 8 | 8 | 7
  Phosphate, Increase to Grade 3: number analyzed (Participants) | 11 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Phosphate, Increase to Grade 3 | 2 | 1 | 3 | 1 | 0 | 2 | 2 | 2 | 3 | 3 | 3 | 0
  Phosphate, Increase to Grade 4: number analyzed (Participants) | 11 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Phosphate, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hypernatremia, Any Grade Increase | 1 | 0 | 1 | 1 | 1 | 2 | 4 | 2 | 1 | 1 | 1 | 2
  Hypernatremia, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hypernatremia, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hypernatremia, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hyponatremia, Any Grade Increase | 4 | 1 | 3 | 3 | 4 | 3 | 3 | 5 | 4 | 4 | 2 | 5
  Hyponatremia, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hyponatremia, Increase to Grade 3 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 1
  Hyponatremia, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Hyponatremia, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urate, Any Grade Increase: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
  Urate, Any Grade Increase | 1 |  | 1 | 1 | 1 | 1 |  | 1 |  |  |  | 1
  Urate, Increase to Grade 3: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
  Urate, Increase to Grade 3 | 0 |  | 0 | 0 | 0 | 0 |  | 0 |  |  |  | 0
  Urate, Increase to Grade 4: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
  Urate, Increase to Grade 4 | 1 |  | 1 | 1 | 1 | 1 |  | 1 |  |  |  | 1
  Hypercalcemia, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 13 | 11 | 12 | 12 | 12 | 12 | 15 | 10 | 16
  Hypercalcemia, Any Grade Increase | 0 | 0 | 2 | 1 | 2 | 2 | 2 | 1 | 3 | 4 | 1 | 1
  Hypercalcemia, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 13 | 11 | 12 | 12 | 12 | 12 | 15 | 10 | 16
  Hypercalcemia, Increase to Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Hypercalcemia, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 13 | 11 | 12 | 12 | 12 | 12 | 15 | 10 | 16
  Hypercalcemia, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypocalcemia, Any Grade Increase: number analyzed (Participants) | 12 | 4 | 13 | 13 | 11 | 12 | 12 | 12 | 12 | 15 | 10 | 16
  Hypocalcemia, Any Grade Increase | 5 | 0 | 4 | 2 | 1 | 3 | 2 | 2 | 5 | 1 | 0 | 3
  Hypocalcemia, Increase to Grade 3: number analyzed (Participants) | 12 | 4 | 13 | 13 | 11 | 12 | 12 | 12 | 12 | 15 | 10 | 16
  Hypocalcemia, Increase to Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypocalcemia, Increase to Grade 4: number analyzed (Participants) | 12 | 4 | 13 | 13 | 11 | 12 | 12 | 12 | 12 | 15 | 10 | 16
  Hypocalcemia, Increase to Grade 4 | 3 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Worst-case Change Post-baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for analysis of following clinical chemistry parameters: Direct Bilirubin (DB), Calcium, Chloride, Carbon Dioxide (CO2), lactate dehydrogenase (LDH) and Protein. The summaries of worst-case change from baseline with respect to normal range was analyzed for only those laboratory tests that were not gradable by CTCAE version 4.03. The number of participants with decreases to low from baseline, changes to normal or no changes from baseline, and increases to high values from baseline have been presented. Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 15 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Participants
  DB, Decrease to Low: number analyzed (Participants) | 10 | 4 | 13 | 13 | 12 | 12 | 12 | 11 | 12 | 18 | 12 | 16
  DB, Decrease to Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DB, Change to Normal or No Change: number analyzed (Participants) | 10 | 4 | 13 | 13 | 12 | 12 | 12 | 11 | 12 | 18 | 12 | 16
  DB, Change to Normal or No Change | 4 | 4 | 9 | 8 | 11 | 8 | 10 | 9 | 9 | 13 | 10 | 14
  DB, Increase to High: number analyzed (Participants) | 10 | 4 | 13 | 13 | 12 | 12 | 12 | 11 | 12 | 18 | 12 | 16
  DB, Increase to High | 6 | 0 | 4 | 5 | 1 | 4 | 2 | 2 | 3 | 5 | 2 | 2
  Calcium, Decrease to Low | 7 | 1 | 7 | 7 | 2 | 6 | 4 | 2 | 5 | 9 | 2 | 5
  Calcium, Change to Normal or No Change | 5 | 3 | 6 | 7 | 8 | 5 | 6 | 10 | 8 | 8 | 6 | 11
  Calcium, Increase to High | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 1 | 2 | 4 | 1
  Chloride, Decrease to Low: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Chloride, Decrease to Low | 1 | 1 | 1 | 3 | 0 | 0 | 1 | 1 | 3 | 3 | 1 | 2
  Chloride, Change to Normal or No Change: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Chloride, Change to Normal or No Change | 5 | 3 | 8 | 10 | 8 | 7 | 5 | 10 | 7 | 9 | 10 | 12
  Chloride, Increase to High: number analyzed (Participants) | 10 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  Chloride, Increase to High | 5 | 0 | 4 | 2 | 4 | 5 | 6 | 1 | 4 | 6 | 1 | 2
  CO2, Decrease to Low: number analyzed (Participants) | 12 | 4 | 13 | 14 | 11 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  CO2, Decrease to Low | 5 | 0 | 5 | 5 | 5 | 3 | 3 | 1 | 5 | 4 | 4 | 2
  CO2, Change to Normal or No Change: number analyzed (Participants) | 12 | 4 | 13 | 14 | 11 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  CO2, Change to Normal or No Change | 7 | 4 | 7 | 7 | 5 | 7 | 9 | 8 | 6 | 14 | 8 | 11
  CO2, Increase to High: number analyzed (Participants) | 12 | 4 | 13 | 14 | 11 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  CO2, Increase to High | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 3 | 2 | 1 | 0 | 3
  Protein, Decrease to Low | 8 | 2 | 5 | 12 | 3 | 7 | 7 | 6 | 7 | 11 | 7 | 10
  Protein, Change to Normal or No Change | 4 | 2 | 8 | 3 | 8 | 5 | 4 | 5 | 5 | 5 | 4 | 5
  Protein, Increase to High | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 1
  LDH, Decrease to Low: number analyzed (Participants) | 11 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  LDH, Decrease to Low | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
  LDH, Change to Normal or No Change: number analyzed (Participants) | 11 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  LDH, Change to Normal or No Change | 5 | 1 | 3 | 6 | 4 | 4 | 3 | 4 | 4 | 1 | 4 | 5
  LDH, Increase to High: number analyzed (Participants) | 11 | 4 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
  LDH, Increase to High | 6 | 3 | 9 | 8 | 8 | 8 | 9 | 7 | 8 | 17 | 8 | 11

9. Primary Outcome: Number of Participants With Worst-case Change Post Baseline Urinalysis Results: Occult Blood and Protein
Description: Urine samples were collected to analyze presence of occult blood and protein in urine by dipstick method. Data for worst-case post baseline urinalysis results is presented. Result for urinalysis parameters were recorded as no change/decreased and increase to trace, 1+, 2+, 3+, >3+ indicating proportional concentrations in the urine sample. Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 10 | 4 | 13 | 13 | 9 | 12 | 12 | 12 | 12 | 18 | 11 | 16
Participants
  Occult Blood, No Change/Decreased: number analyzed (Participants) | 10 | 4 | 13 | 13 | 9 | 12 | 12 | 12 | 11 | 18 | 11 | 16
  Occult Blood, No Change/Decreased | 5 | 2 | 6 | 6 | 6 | 8 | 6 | 9 | 4 | 11 | 7 | 12
  Occult Blood, Increase to TRACE: number analyzed (Participants) | 10 | 4 | 13 | 13 | 9 | 12 | 12 | 12 | 11 | 18 | 11 | 16
  Occult Blood, Increase to TRACE | 1 | 2 | 3 | 4 | 0 | 2 | 2 | 1 | 5 | 1 | 0 | 0
  Occult Blood, Increase to 1+: number analyzed (Participants) | 10 | 4 | 13 | 13 | 9 | 12 | 12 | 12 | 11 | 18 | 11 | 16
  Occult Blood, Increase to 1+ | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 4 | 2 | 3
  Occult Blood, Increase to 2+: number analyzed (Participants) | 10 | 4 | 13 | 13 | 9 | 12 | 12 | 12 | 11 | 18 | 11 | 16
  Occult Blood, Increase to 2+ | 3 | 0 | 2 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 2 | 1
  Occult Blood, Increase to 3+: number analyzed (Participants) | 10 | 4 | 13 | 13 | 9 | 12 | 12 | 12 | 11 | 18 | 11 | 16
  Occult Blood, Increase to 3+ | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
  Occult Blood, Increase to >3+: number analyzed (Participants) | 10 | 4 | 13 | 13 | 9 | 12 | 12 | 12 | 11 | 18 | 11 | 16
  Occult Blood, Increase to >3+ | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Protein, No Change/Decreased | 5 | 2 | 7 | 3 | 2 | 5 | 5 | 6 | 5 | 8 | 4 | 5
  Protein, Increase to TRACE | 2 | 0 | 1 | 6 | 1 | 2 | 2 | 2 | 1 | 2 | 0 | 1
  Protein, Increase to 1+ | 1 | 0 | 3 | 0 | 2 | 2 | 4 | 2 | 2 | 4 | 2 | 6
  Protein, Increase to 2+ | 2 | 0 | 2 | 3 | 2 | 0 | 1 | 2 | 2 | 2 | 2 | 3
  Protein, Increase to 3+ | 0 | 2 | 0 | 1 | 1 | 3 | 0 | 0 | 2 | 2 | 3 | 1
  Protein, Increase to >3+ | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Change From Baseline in Urine Potential of Hydrogen (pH)
Description: Urine samples were collected to analyze urine pH levels. Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Potential of Hydrogen (pH)
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 10 | 4 | 13 | 12 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Potential of Hydrogen (pH)
  Baseline (Day 1) | 5.9 (0.46) | 5.8 (0.65) | 6.0 (0.90) | 5.8 (0.69) | 6.1 (0.68) | 5.8 (0.62) | 6.4 (0.87) | 5.6 (0.48) | 5.9 (0.82) | 6.1 (0.82) | 5.9 (1.18) | 5.7 (0.70)
  Change from baseline (up to approx. 4.5 years): number analyzed (Participants) | 5 | 3 | 7 | 3 | 6 | 5 | 3 | 9 | 4 | 13 | 5 | 12
  Change from baseline (up to approx. 4.5 years) | 0.1 (1.08) | -0.2 (0.76) | 0.4 (1.38) | 0.2 (0.29) | -0.3 (0.61) | 0.6 (0.42) | -0.5 (0.50) | 0.2 (0.66) | 0.4 (1.03) | 0.2 (0.80) | 0.4 (0.55) | 0.2 (1.05)

11. Primary Outcome: Change From Baseline in Urine Specific Gravity
Description: Urine samples were collected to analyze urine specific gravity using dipstick method. Baseline (Day 1) was defined as latest pre-dose assessment with a non-missing value, including unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 7 | 4 | 13 | 11 | 6 | 12 | 9 | 11 | 12 | 18 | 11 | 14
Ratio
  Baseline (Day 1) | 1.0217 (0.00687) | 1.0253 (0.00660) | 1.0169 (0.00946) | 1.0175 (0.00682) | 1.0217 (0.00931) | 1.0175 (0.00544) | 1.0133 (0.00661) | 1.0167 (0.00736) | 1.0193 (0.00612) | 1.0152 (0.00817) | 1.0174 (0.00713) | 1.0139 (0.00627)
  Change from baseline (up to approx. 4.5 years): number analyzed (Participants) | 3 | 3 | 7 | 3 | 2 | 5 | 2 | 7 | 3 | 13 | 5 | 10
  Change from baseline (up to approx. 4.5 years) | 0.0003 (0.00058) | -0.0090 (0.01217) | -0.0013 (0.01072) | 0.0023 (0.00643) | 0.0075 (0.00354) | -0.0020 (0.00671) | 0.0050 (0.00707) | 0.0029 (0.01029) | -0.0010 (0.00529) | 0.0005 (0.00782) | -0.0026 (0.00792) | 0.0067 (0.00830)

12. Primary Outcome: Change From Baseline in Vital Signs: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: Blood pressures (DBP and SBP) were measured after resting for at least 5 minutes in a supine or semi-recumbent position. Baseline (Day 1) was defined as latest pre-dose assessment with a non-missing value, including unscheduled visits. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All treated population. Data was not collected where number of participants analyzed is 0. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16 | 12 | 12 | 12 | 12 | 13 | 17 | 12 | 16
Millimeters of mercury (mmHg)
  DBP, BASELINE (Day 1) | 72.3 (7.67) | 86.0 (12.49) | 79.5 (9.36) | 71.4 (12.04) | 73.6 (17.15) | 75.1 (9.08) | 78.4 (11.13) | 76.1 (7.14) | 72.2 (8.52) | 74.9 (8.77) | 72.9 (11.85) | 77.8 (10.61)
  DBP, WEEK 79 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
  DBP, WEEK 79 DAY 1, Predose |  |  |  |  | -5.0 | 3.0 |  |  | 19.0 | 2.0 | -1.0 | -23.0
  DBP, WEEK 79 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
  DBP, WEEK 79 DAY 1, 0.25hour Post-Dose |  |  |  |  | -8.0 | -3.0 |  |  | 12.0 | -2.0 | -11.0 | -14.0
  DBP, WEEK 79 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
  DBP, WEEK 79 DAY 1, 1hour Post-Dose |  |  |  |  | -5.0 | -6.0 |  |  | 19.0 | 5.0 | -10.0 | -44.0
  DBP, WEEK 91 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  DBP, WEEK 91 DAY 1, Predose |  |  |  |  |  | 6.0 |  | 4.0 | -4.0 | -26.0 |  |
  DBP, WEEK 91 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  DBP, WEEK 91 DAY 1, 0.25hour Post-Dose |  |  |  |  |  | 0.0 (0.0) |  | 10.0 | 1.0 | -15.0 |  |
  DBP, WEEK 91 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  DBP, WEEK 91 DAY 1, 1hour Post-Dose |  |  |  |  |  | 10.0 |  | 3.0 | -2.0 | -16.0 |  |
  DBP, WEEK 94 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  DBP, WEEK 94 DAY 1, Predose |  |  |  |  |  |  | -24.0 |  | 4.0 | -7.0 | -2.0 |
  DBP, WEEK 94 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  DBP, WEEK 94 DAY 1, 0.25hour Post-Dose |  |  |  |  |  |  | -21.0 |  | 6.0 | 4.0 | 3.0 |
  DBP, WEEK 94 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  DBP, WEEK 94 DAY 1, 1hour Post-Dose |  |  |  |  |  |  | -21.0 |  | 14.0 | -5.0 | 2.0 |
  DBP, WEEK 109 DAY 1, Predose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
  DBP, WEEK 109 DAY 1, Predose | 5.0 |  | 2.0 | -1.7 (2.08) |  |  |  |  | -4.5 (0.71) | 6.0 |  | -14.0
  DBP, WEEK 109 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
  DBP, WEEK 109 DAY 1, 0.25hour Post-Dose | -4.0 |  | -2.0 | 0.0 (6.24) |  |  |  |  | 1.5 (7.78) | 6.0 |  | -21.0
  DBP, WEEK 109 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
  DBP, WEEK 109 DAY 1, 1hour Post-Dose | 9.0 |  | 2.0 | 0.0 (5.57) |  |  |  |  | 5.5 (2.12) | 3.0 |  | -27.0
  DBP, WEEK 133 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  DBP, WEEK 133 DAY 1, Predose |  |  |  | -2.0 (2.83) |  |  |  |  | 6.0 |  |  | -16.0
  DBP, WEEK 133 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  DBP, WEEK 133 DAY 1, 0.25hour Post-Dose |  |  |  | 1.0 (7.07) |  |  |  |  | 3.0 |  |  | -18.0
  DBP, WEEK 133 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  DBP, WEEK 133 DAY 1, 1hour Post-Dose |  |  |  | 4.5 (3.54) |  |  |  |  | 8.0 |  |  | -14.0
  DBP, WEEK 153 DAY 8, Predose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, WEEK 153 DAY 8, Predose |  |  | 5.0 |  |  |  |  |  |  |  |  |
  DBP, WEEK 153 DAY 8, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, WEEK 153 DAY 8, 0.25hour Post-Dose |  |  | 10.0 |  |  |  |  |  |  |  |  |
  DBP, WEEK 153 DAY 8, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, WEEK 153 DAY 8, 1hour Post-Dose |  |  | 4.0 |  |  |  |  |  |  |  |  |
  DBP, WEEK 169 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  DBP, WEEK 169 DAY 1, Predose |  |  |  |  |  |  |  |  | 11.0 | -16.5 (26.16) |  |
  DBP, WEEK 169 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  DBP, WEEK 169 DAY 1, 0.25hour Post-Dose |  |  |  |  |  |  |  |  | 6.0 | 3.0 (4.24) |  |
  DBP, WEEK 169 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  DBP, WEEK 169 DAY 1, 1hour Post-Dose |  |  |  |  |  |  |  |  | 7.0 | -11.0 (16.97) |  |
  DBP, WEEK 169 DAY 8, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  DBP, WEEK 169 DAY 8, Predose |  |  |  |  |  |  |  |  | 11.0 |  |  |
  DBP, WEEK 169 DAY 8, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  DBP, WEEK 169 DAY 8, 0.25hour Post-Dose |  |  |  |  |  |  |  |  | 6.0 |  |  |
  DBP, WEEK 169 DAY 8, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  DBP, WEEK 169 DAY 8, 1hour Post-Dose |  |  |  |  |  |  |  |  | -5.0 |  |  |
  DBP, WEEK 173 DAY 1, Predose: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, WEEK 173 DAY 1, Predose |  | -14.0 |  |  |  |  |  |  |  |  |  |
  DBP, WEEK 173 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, WEEK 173 DAY 1, 0.25hour Post-Dose |  | -10.0 |  |  |  |  |  |  |  |  |  |
  DBP, WEEK 173 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, WEEK 173 DAY 1, 1hour Post-Dose |  | -3.0 |  |  |  |  |  |  |  |  |  |
  DBP, WEEK 221 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, WEEK 221 DAY 1, Predose |  |  |  | -2.0 |  |  |  |  |  |  |  |
  DBP, WEEK 221 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, WEEK 221 DAY 1, 0.25hour Post-Dose |  |  |  | -10.0 |  |  |  |  |  |  |  |
  DBP, WEEK 221 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, WEEK 221 DAY 1, 1hour Post-Dose |  |  |  | 2.0 |  |  |  |  |  |  |  |
  SBP, BASELINE (Day 1) | 127.8 (18.62) | 137.5 (7.05) | 136.1 (26.03) | 125.3 (15.71) | 136.4 (18.99) | 129.7 (15.13) | 132.8 (17.88) | 135.4 (16.68) | 122.3 (13.94) | 143.3 (25.93) | 126.8 (21.48) | 138.5 (21.29)
  SBP, WEEK 79 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
  SBP, WEEK 79 DAY 1, Predose |  |  |  |  | 11.0 | 5.0 |  |  | 8.0 | 16.0 | -17.0 | -21.0
  SBP, WEEK 79 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
  SBP, WEEK 79 DAY 1, 0.25hour Post-Dose |  |  |  |  | 10.0 | -3.0 |  |  | 8.0 | 9.0 | -36.0 | -7.0
  SBP, WEEK 79 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
  SBP, WEEK 79 DAY 1, 1hour Post-Dose |  |  |  |  | 12.0 | -2.0 |  |  | -1.0 | 0.0 (0.0) | -41.0 | -1.0
  SBP, WEEK 91 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  SBP, WEEK 91 DAY 1, Predose |  |  |  |  |  | -5.0 |  | -2.0 | 4.0 | -22.0 |  |
  SBP, WEEK 91 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  SBP, WEEK 91 DAY 1, 0.25hour Post-Dose |  |  |  |  |  | -15.0 |  | 17.0 | 12.0 | -31.0 |  |
  SBP, WEEK 91 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  SBP, WEEK 91 DAY 1, 1hour Post-Dose |  |  |  |  |  | 21.0 |  | 16.0 | 4.0 | -15.0 |  |
  SBP, WEEK 94 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  SBP, WEEK 94 DAY 1, Predose |  |  |  |  |  |  | -28.0 |  | -5.0 | -38.0 | 12.0 |
  SBP, WEEK 94 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  SBP, WEEK 94 DAY 1, 0.25hour Post-Dose |  |  |  |  |  |  | -30.0 |  | -4.0 | -23.0 | 3.0 |
  SBP, WEEK 94 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  SBP, WEEK 94 DAY 1, 1hour Post-Dose |  |  |  |  |  |  | -35.0 |  | -4.0 | -32.0 | -5.0 |
  SBP, WEEK 109 DAY 1, Predose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
  SBP, WEEK 109 DAY 1, Predose | 9.0 |  | -1.0 | -4.7 (16.01) |  |  |  |  | -1.0 (5.66) | -11.0 |  | -22.0
  SBP, WEEK 109 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
  SBP, WEEK 109 DAY 1, 0.25hour Post-Dose | 3.0 |  | 1.0 | 1.3 (15.89) |  |  |  |  | -7.5 (0.71) | 0.0 (0.0) |  | -23.0
  SBP, WEEK 109 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
  SBP, WEEK 109 DAY 1, 1hour Post-Dose | 3.0 |  | -3.0 | 7.3 (16.56) |  |  |  |  | -1.5 (4.95) | 8.0 |  | -31.0
  SBP, WEEK 133 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  SBP, WEEK 133 DAY 1, Predose |  |  |  | -9.0 (1.41) |  |  |  |  | 4.0 |  |  | -16.0
  SBP, WEEK 133 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  SBP, WEEK 133 DAY 1, 0.25hour Post-Dose |  |  |  | 3.0 (9.90) |  |  |  |  | -3.0 |  |  | -2.0
  SBP, WEEK 133 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  SBP, WEEK 133 DAY 1, 1hour Post-Dose |  |  |  | 5.0 (19.80) |  |  |  |  | -1.0 |  |  | -1.0
  SBP, WEEK 153 DAY 8, Predose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, WEEK 153 DAY 8, Predose |  |  | -3.0 |  |  |  |  |  |  |  |  |
  SBP, WEEK 153 DAY 8, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, WEEK 153 DAY 8, 0.25hour Post-Dose |  |  | 13.0 |  |  |  |  |  |  |  |  |
  SBP, WEEK 153 DAY 8, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, WEEK 153 DAY 8, 1hour Post-Dose |  |  | 7.0 |  |  |  |  |  |  |  |  |
  SBP, WEEK 169 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  SBP, WEEK 169 DAY 1, Predose |  |  |  |  |  |  |  |  | -5.0 | -16.5 (28.99) |  |
  SBP, WEEK 169 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  SBP, WEEK 169 DAY 1, 0.25hour Post-Dose |  |  |  |  |  |  |  |  | -5.0 | -9.5 (7.78) |  |
  SBP, WEEK 169 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  SBP, WEEK 169 DAY 1, 1hour Post-Dose |  |  |  |  |  |  |  |  | -1.0 | -6.5 (9.19) |  |
  SBP, WEEK 169 DAY 8, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  SBP, WEEK 169 DAY 8, Predose |  |  |  |  |  |  |  |  | 10.0 |  |  |
  SBP, WEEK 169 DAY 8, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  SBP, WEEK 169 DAY 8, 0.25hour Post-Dose |  |  |  |  |  |  |  |  | 11.0 |  |  |
  SBP, WEEK 169 DAY 8, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  SBP, WEEK 169 DAY 8, 1hour Post-Dose |  |  |  |  |  |  |  |  | 17.0 |  |  |
  SBP, WEEK 173 DAY 1, Predose: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, WEEK 173 DAY 1, Predose |  | -7.0 |  |  |  |  |  |  |  |  |  |
  SBP, WEEK 173 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, WEEK 173 DAY 1, 0.25hour Post-Dose |  | -7.0 |  |  |  |  |  |  |  |  |  |
  SBP, WEEK 173 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, WEEK 173 DAY 1, 1hour Post-Dose |  | -5.0 |  |  |  |  |  |  |  |  |  |
  SBP, WEEK 221 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, WEEK 221 DAY 1, Predose |  |  |  | 18.0 |  |  |  |  |  |  |  |
  SBP, WEEK 221 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, WEEK 221 DAY 1, 0.25hour Post-Dose |  |  |  | 15.0 |  |  |  |  |  |  |  |
  SBP, WEEK 221 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, WEEK 221 DAY 1, 1hour Post-Dose |  |  |  | 32.0 |  |  |  |  |  |  |  |

13. Primary Outcome: Change From Baseline in Vital Signs : Pulse Rate
Description: Pulse rate was measured after resting for at least 5 minutes in a supine or semi-recumbent position. Baseline (Day 1) was defined as latest pre-dose assessment with a non-missing value, including unscheduled visits. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16 | 12 | 12 | 12 | 12 | 13 | 17 | 12 | 16
beats per minute
  BASELINE (Day 1) | 72.8 (9.01) | 73.8 (11.90) | 76.0 (17.10) | 72.8 (14.65) | 73.7 (13.05) | 76.2 (12.69) | 75.5 (11.21) | 79.6 (13.36) | 73.3 (14.31) | 74.1 (10.76) | 81.0 (10.05) | 75.3 (10.82)
  WEEK 79 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
  WEEK 79 DAY 1, Predose |  |  |  |  | -9.0 | -18.0 |  |  | -14.0 | 9.0 | 1.0 | 4.0
  WEEK 79 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
  WEEK 79 DAY 1, 0.25hour Post-Dose |  |  |  |  | -6.0 | -6.0 |  |  | 6.0 | -2.0 | 2.0 | -9.0
  WEEK 79 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
  WEEK 79 DAY 1, 1hour Post-Dose |  |  |  |  | -18.0 | 6.0 |  |  | 13.0 | -2.0 | 4.0 | -6.0
  WEEK 91 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  WEEK 91 DAY 1, Predose |  |  |  |  |  | 1.0 |  | -5.0 | 24.0 | -5.0 |  |
  WEEK 91 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  WEEK 91 DAY 1, 0.25hour Post-Dose |  |  |  |  |  | -2.0 |  | -19.0 | 12.0 | -9.0 |  |
  WEEK 91 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  WEEK 91 DAY 1, 1hour Post-Dose |  |  |  |  |  | -6.0 |  | -11.0 | 11.0 | -19.0 |  |
  WEEK 94 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  WEEK 94 DAY 1, Predose |  |  |  |  |  |  | -5.0 |  | -14.0 | 21.0 | 13.0 |
  WEEK 94 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  WEEK 94 DAY 1, 0.25hour Post-Dose |  |  |  |  |  |  | -4.0 |  | -22.0 | 16.0 | 12.0 |
  WEEK 94 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  WEEK 94 DAY 1, 1hour Post-Dose |  |  |  |  |  |  | -4.0 |  | -28.0 | 11.0 | 14.0 |
  WEEK 109 DAY 1, Predose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
  WEEK 109 DAY 1, Predose | -19.0 |  | -22.0 | 8.3 (5.13) |  |  |  |  | -6.0 (8.49) | -12.0 |  | -9.0
  WEEK 109 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
  WEEK 109 DAY 1, 0.25hour Post-Dose | -18.0 |  | -24.0 | 0.3 (3.06) |  |  |  |  | 10.5 (41.72) | -16.0 |  | -8.0
  WEEK 109 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
  WEEK 109 DAY 1, 1hour Post-Dose | -4.0 |  | -25.0 | 1.3 (5.69) |  |  |  |  | -8.0 (11.31) | -12.0 |  | 0.0
  WEEK 133 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  WEEK 133 DAY 1, Predose |  |  |  | 6.5 (9.19) |  |  |  |  | -11.0 |  |  | -5.0
  WEEK 133 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  WEEK 133 DAY 1, 0.25hour Post-Dose |  |  |  | 4.5 (0.71) |  |  |  |  | -12.0 |  |  | -5.0
  WEEK 133 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  WEEK 133 DAY 1, 1hour Post-Dose |  |  |  | 5.5 (2.12) |  |  |  |  | -16.0 |  |  | -17.0
  WEEK 153 DAY 8, Predose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 153 DAY 8, Predose |  |  | -8.0 |  |  |  |  |  |  |  |  |
  WEEK 153 DAY 8, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 153 DAY 8, 0.25hour Post-Dose |  |  | -10.0 |  |  |  |  |  |  |  |  |
  WEEK 153 DAY 8, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 153 DAY 8, 1hour Post-Dose |  |  | -9.0 |  |  |  |  |  |  |  |  |
  WEEK 169 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  WEEK 169 DAY 1, Predose |  |  |  |  |  |  |  |  | -15.0 | -21.0 (5.66) |  |
  WEEK 169 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  WEEK 169 DAY 1, 0.25hour Post-Dose |  |  |  |  |  |  |  |  | -23.0 | -19.0 (2.83) |  |
  WEEK 169 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  WEEK 169 DAY 1, 1hour Post-Dose |  |  |  |  |  |  |  |  | -20.0 | -21.0 (1.41) |  |
  WEEK 169 DAY 8, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WEEK 169 DAY 8, Predose |  |  |  |  |  |  |  |  | -21.0 |  |  |
  WEEK 169 DAY 8, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WEEK 169 DAY 8, 0.25hour Post-Dose |  |  |  |  |  |  |  |  | -17.0 |  |  |
  WEEK 169 DAY 8, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WEEK 169 DAY 8, 1hour Post-Dose |  |  |  |  |  |  |  |  | -20.0 |  |  |
  WEEK 173 DAY 1, Predose: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 173 DAY 1, Predose |  | -7.0 |  |  |  |  |  |  |  |  |  |
  WEEK 173 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 173 DAY 1, 0.25hour Post-Dose |  | -5.0 |  |  |  |  |  |  |  |  |  |
  WEEK 173 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 173 DAY 1, 1hour Post-Dose |  | -8.0 |  |  |  |  |  |  |  |  |  |
  WEEK 221 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 221 DAY 1, Predose |  |  |  | -4.0 |  |  |  |  |  |  |  |
  WEEK 221 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 221 DAY 1, 0.25hour Post-Dose |  |  |  | 2.0 |  |  |  |  |  |  |  |
  WEEK 221 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 221 DAY 1, 1hour Post-Dose |  |  |  | 8.0 |  |  |  |  |  |  |  |

14. Primary Outcome: Change From Baseline in Vital Signs : Temperature
Description: Temperature was measured after resting for at least 5 minutes in a supine or semi-recumbent position. Baseline (Day 1) was defined as latest pre-dose assessment with a non-missing value, including unscheduled visits. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Degree Celsius (C)
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16 | 12 | 12 | 12 | 12 | 13 | 17 | 12 | 16
Degree Celsius (C)
  BASELINE (Day 1) | 36.61 (0.417) | 36.70 (0.346) | 36.46 (0.307) | 36.43 (0.334) | 36.46 (0.348) | 36.44 (0.291) | 36.52 (0.432) | 36.68 (0.305) | 36.53 (0.338) | 36.48 (0.571) | 36.51 (0.581) | 36.58 (0.397)
  WEEK 79 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
  WEEK 79 DAY 1, Predose |  |  |  |  | -0.30 | 0.10 |  |  | 0.70 | -0.10 | 1.30 | 0.00 (0.00)
  WEEK 79 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
  WEEK 79 DAY 1, 0.25hour Post-Dose |  |  |  |  | -0.30 | 0.10 |  |  | -0.20 | -0.10 | 1.60 | 0.00 (0.00)
  WEEK 79 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
  WEEK 79 DAY 1, 1hour Post-Dose |  |  |  |  | -0.10 | 0.40 |  |  | 0.50 | 0.00 (0.00) | 1.40 | 0.00 (0.00)
  WEEK 91 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  WEEK 91 DAY 1, Predose |  |  |  |  |  | 0.40 |  | -0.60 | 0.50 | -0.70 |  |
  WEEK 91 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  WEEK 91 DAY 1, 0.25hour Post-Dose |  |  |  |  |  | 0.40 |  | -0.80 | 0.10 | 0.20 |  |
  WEEK 91 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  WEEK 91 DAY 1, 1hour Post-Dose |  |  |  |  |  | 0.50 |  | -0.50 | 0.50 | 0.30 |  |
  WEEK 94 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  WEEK 94 DAY 1, Predose |  |  |  |  |  |  | -0.20 |  | 0.10 | -0.30 | 0.30 |
  WEEK 94 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  WEEK 94 DAY 1, 0.25hour Post-Dose |  |  |  |  |  |  | -0.30 |  | 0.30 | 0.10 | 0.30 |
  WEEK 94 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  WEEK 94 DAY 1, 1hour Post-Dose |  |  |  |  |  |  | -0.40 |  | 0.00 (0.00) | 0.10 | 0.30 |
  WEEK 109 DAY 1, Predose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
  WEEK 109 DAY 1, Predose | -0.90 |  | -0.80 | 0.20 (0.173) |  |  |  |  | 0.20 (0.283) | -0.20 |  | 0.40
  WEEK 109 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
  WEEK 109 DAY 1, 0.25hour Post-Dose | -1.20 |  | -0.80 | 0.07 (0.153) |  |  |  |  | 0.15 (0.071) | 0.20 |  | 0.40
  WEEK 109 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
  WEEK 109 DAY 1, 1hour Post-Dose | -1.20 |  | -0.50 | 0.10 (0.173) |  |  |  |  | 0.15 (0.071) | 0.10 |  | 0.40
  WEEK 133 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  WEEK 133 DAY 1, Predose |  |  |  | 0.60 (0.283) |  |  |  |  | 0.40 |  |  | 1.00
  WEEK 133 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  WEEK 133 DAY 1, 0.25hour Post-Dose |  |  |  | 0.25 (0.071) |  |  |  |  | 0.30 |  |  | 0.70
  WEEK 133 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  WEEK 133 DAY 1, 1hour Post-Dose |  |  |  | 0.45 (0.071) |  |  |  |  | 0.10 |  |  | 0.20
  WEEK 148 DAY 8, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WEEK 148 DAY 8, Predose |  |  |  |  |  |  |  |  |  |  | 0.00 |
  WEEK 148 DAY 8, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WEEK 148 DAY 8, 0.25hour Post-Dose |  |  |  |  |  |  |  |  |  |  | -0.30 |
  WEEK 148 DAY 8, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WEEK 148 DAY 8, 1hour Post-Dose |  |  |  |  |  |  |  |  |  |  | -0.30 |
  WEEK 153 DAY 8, Predose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 153 DAY 8, Predose |  |  | 0.20 |  |  |  |  |  |  |  |  |
  WEEK 153 DAY 8, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 153 DAY 8, 0.25hour Post-Dose |  |  | -0.10 |  |  |  |  |  |  |  |  |
  WEEK 153 DAY 8, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 153 DAY 8, 1hour Post-Dose |  |  | 0.00 (0.00) |  |  |  |  |  |  |  |  |
  WEEK 169 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  WEEK 169 DAY 1, Predose |  |  |  |  |  |  |  |  | -0.20 | 0.10 |  |
  WEEK 169 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  WEEK 169 DAY 1, 0.25hour Post-Dose |  |  |  |  |  |  |  |  | 0.10 | 0.05 (0.636) |  |
  WEEK 169 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  WEEK 169 DAY 1, 1hour Post-Dose |  |  |  |  |  |  |  |  | 0.10 | -0.05 (0.071) |  |
  WEEK 169 DAY 8, Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WEEK 169 DAY 8, Predose |  |  |  |  |  |  |  |  | -0.20 |  |  |
  WEEK 169 DAY 8, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WEEK 169 DAY 8, 0.25hour Post-Dose |  |  |  |  |  |  |  |  | 0.40 |  |  |
  WEEK 169 DAY 8, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WEEK 169 DAY 8, 1hour Post-Dose |  |  |  |  |  |  |  |  | -0.30 |  |  |
  WEEK 173 DAY 1, Predose: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 173 DAY 1, Predose |  | -0.30 |  |  |  |  |  |  |  |  |  |
  WEEK 173 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 173 DAY 1, 0.25hour Post-Dose |  | -0.40 |  |  |  |  |  |  |  |  |  |
  WEEK 173 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 173 DAY 1, 1hour Post-Dose |  | -0.40 |  |  |  |  |  |  |  |  |  |
  WEEK 221 DAY 1, Predose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 221 DAY 1, Predose |  |  |  | -0.10 |  |  |  |  |  |  |  |
  WEEK 221 DAY 1, 0.25hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 221 DAY 1, 0.25hour Post-Dose |  |  |  | -0.10 |  |  |  |  |  |  |  |
  WEEK 221 DAY 1, 1hour Post-Dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WEEK 221 DAY 1, 1hour Post-Dose |  |  |  | -0.20 |  |  |  |  |  |  |  |

15. Primary Outcome: Overall Response Rate (ORR) as Defined by the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma (MM)
Description: ORR was defined as the percentage of participants with a confirmed partial response (PR) or better (i.e., PR, very good partial response [VGPR], complete response [CR] and stringent complete response [sCR]), according to the International Myeloma Working Group (IMWG) Response Criteria. CR: negative immunofixation of serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasmacytomas in the bone marrow; sCR: stringent complete response, CR as above plus normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR: serum and urine M-component detectable by immunofixation but not on electrophoresis OR >= 90% reduction in serum M-component plus urine M-component <100 mg/24 h; PR: >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200 mg/24 h. Confidence intervals were based on the exact method.
Time Frame: Up to approximately 4.5 years
Population: All treated population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Percentage of Participants | 58 [27.7 to 84.8] | 75 [19.4 to 99.4] | 69 [38.6 to 90.9] | 69 [41.3 to 89.0] | 50 [21.1 to 78.9] | 83 [51.6 to 97.9] | 92 [61.5 to 99.8] | 75 [42.8 to 94.5] | 62 [31.6 to 86.1] | 78 [52.4 to 93.6] | 50 [21.1 to 78.9] | 69 [41.3 to 89.0]

16. Secondary Outcome: Maximum Observed Concentration (Cmax) for Belantamab Mafodotin Antibody-drug Conjugate (ADC), Treatment A
Description: Blood samples were collected at indicated timepoints for pharmacokinetic (PK) analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0, 2 and 24 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: Pharmacokinetic (PK) population included all participants in all treated population from whom at least one PK sample was obtained, analyzed, and was measurable. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/ millilitre (ug/mL)
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 15
Microgram/ millilitre (ug/mL)
  CYCLE 1 DAY 1 | 43.58 (21.78) | 36.41 (17.06) | 25.22 (16.53) | 39.99 (25.03)
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 12 | 0
  CYCLE 1 DAY 8 |  |  | 27.60 (16.27) |

17. Secondary Outcome: Area Under the Concentration Time Curve (AUC) From Time 0 to 504 Hours (0-504h) for Belantamab Mafodotin ADC, Treatment A
Description: Blood samples were collected at indicated timepoints for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1; Cycle 1 Day 4; Cycle 1 Day 8; Cycle 1 Day 11; Cycle 1 Day 15-21
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram/millilitre (h*ug/mL)
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 4 | 3 | 9 | 9
Hour*microgram/millilitre (h*ug/mL) | 3848.41 (24.25) | 4802.83 (34.51) | 4365.82 (10.25) | 4127.66 (17.98)

18. Secondary Outcome: AUC (0-672h) for Belantamab Mafodotin ADC, Treatment A
Description: as for outcome 17
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1; Cycle 1 Day 4; Cycle 1 Day 8; Cycle 1 Day 11; Cycle 1 Day 15-21; Cycle 1 Day 28
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 4 | 3 | 9 | 9
h*ug/mL | 4093.12 (24.45) | 5114.28 (34.72) | 4699.00 (11.10) | 4432.11 (17.65)

19. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) for Belantamab Mafodotin ADC, Treatment A
Description: as for outcome 17
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 17
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 15
Hour
  CYCLE 1 DAY 1 | 2.050 [0.57 to 2.37] | 1.342 [0.50 to 2.17] | 1.100 [0.57 to 2.20] | 2.000 [0.53 to 2.42]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 12 | 0
  CYCLE 1 DAY 8 |  |  | 1.108 [0.57 to 23.93] |

20. Secondary Outcome: Time of Last Observed Quantifiable Concentration (Tlast) for Belantamab Mafodotin ADC, Treatment A
Description: Blood samples were collected at indicated timepoints for PK analysis. PK parameter was determined using standard non-compartmental methods. Tlast is the time of last observed quantifiable concentration of belantamab mafodotin in Cycle 1 which extended beyond protocol defined duration for some participants across treatment groups.
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1 and Cycle 1 Day 4; Cycle 1 Day 8; Cycle 1 Day 11; Cycle 1 Day 15-21; Cycle 1 Day 29; pre-dose Cycle 2 Day 28
Population: Pharmacokinetic (PK) population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16
Hour | 181.467 [25.50 to 698.22] | 685.608 [191.58 to 697.75] | 674.833 [94.40 to 1273.75] | 671.717 [2.00 to 1342.83]

21. Secondary Outcome: Trough Concentration Prior to the Next Dose for Each Cycle (Ctrough) for Belantamab Mafodotin ADC, Treatment A
Description: as for outcome 17
Time Frame: Cycle 1: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Days 1 and 8; Weeks 5, 9, and 13: Pre-Dose and Post-Dose on Days 1 and 8
Population: Pharmacokinetic (PK) population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 1 | 3 | 12 | 11
ug/mL
  CYCLE 1 DAY 1: number analyzed (Participants) | 0 | 3 | 12 | 11
  CYCLE 1 DAY 1 |  | 1.79 [0.7 to 1.8] | 3.52 [2.5 to 4.7] | 1.08 [0.7 to 1.5]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 10 | 0
  CYCLE 1 DAY 8 |  |  | 1.30 [0.7 to 2.4] |
  WEEK 5 DAY 1: number analyzed (Participants) | 0 | 2 | 9 | 2
  WEEK 5 DAY 1 |  | NA [0.5 to 2.6] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 5.05 [2.4 to 7.0] | NA [0.6 to 1.0] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  WEEK 5 DAY 8: number analyzed (Participants) | 0 | 0 | 8 | 0
  WEEK 5 DAY 8 |  |  | 1.17 [0.1 to 3.6] |
  WEEK 9 DAY 1: number analyzed (Participants) | 0 | 1 | 7 | 2
  WEEK 9 DAY 1 |  | NA [2.3 to 2.3] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 4.89 [3.0 to 8.4] | NA [2.3 to 2.9] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  WEEK 9 DAY 8: number analyzed (Participants) | 0 | 0 | 3 | 0
  WEEK 9 DAY 8 |  |  | 2.03 [1.8 to 3.9] |
  WEEK 13 DAY 1: number analyzed (Participants) | 1 | 0 | 2 | 2
  WEEK 13 DAY 1 | NA [0.7 to 0.7] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [4.4 to 6.5] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [2.3 to 3.5] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  WEEK 13 DAY 8: number analyzed (Participants) | 0 | 0 | 1 | 0
  WEEK 13 DAY 8 |  |  | NA [1.6 to 1.6] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |

22. Secondary Outcome: Observed Plasma Concentration at the End of Infusion (C-EOI) for Belantamab Mafodotin ADC, Treatment A
Description: as for outcome 17
Time Frame: Cycle 1: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Days 1 and Day 8; Weeks 5, 9, and 13: Pre-Dose and Post-Dose on Days 1 and 8
Population: as for outcome 17
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 11 | 4 | 12 | 15
ug/mL
  CYCLE 1 DAY 1 | 39.10 [27.2 to 49.5] | 36.05 [29.6 to 44.5] | 25.05 [18.2 to 31.5] | 41.80 [14.0 to 51.3]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 12 | 0
  CYCLE 1 DAY 8 |  |  | 26.55 [18.6 to 35.2] |
  WEEK 5 DAY 1: number analyzed (Participants) | 0 | 4 | 10 | 10
  WEEK 5 DAY 1 |  | 35.45 [33.8 to 42.0] | 23.00 [20.5 to 27.2] | 36.75 [25.6 to 96.2]
  WEEK 5 DAY 8: number analyzed (Participants) | 0 | 0 | 9 | 0
  WEEK 5 DAY 8 |  |  | 27.10 [23.6 to 41.8] |
  WEEK 9 DAY 1: number analyzed (Participants) | 6 | 1 | 8 | 2
  WEEK 9 DAY 1 | 42.35 [31.1 to 49.5] | NA [34.5 to 34.5] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 23.50 [15.3 to 31.8] | NA [30.4 to 55.5] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  WEEK 9 DAY 8: number analyzed (Participants) | 0 | 0 | 6 | 0
  WEEK 9 DAY 8 |  |  | 25.60 [17.1 to 31.1] |
  WEEK 13 DAY 1: number analyzed (Participants) | 1 | 0 | 2 | 5
  WEEK 13 DAY 1 | NA [27.1 to 27.1] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [16.8 to 31.6] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 38.40 [28.1 to 50.9]
  WEEK 13 DAY 8: number analyzed (Participants) | 0 | 0 | 2 | 0
  WEEK 13 DAY 8 |  |  | NA [21.7 to 30.2] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |

23. Secondary Outcome: Cmax for Belantamab Mafodotin ADC, Treatment B
Description: as for outcome 17
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
ug/mL
  CYCLE 1 DAY 1: number analyzed (Participants) | 12 | 12 | 12 | 12 | 13 | 18 | 11 | 16
  CYCLE 1 DAY 1 | 52.24 (31.87) | 49.50 (21.38) | 61.16 (36.74) | 51.29 (26.03) | 21.34 (34.67) | 46.95 (23.24) | 27.79 (37.28) | 64.00 (38.60)
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 0 | 12 | 0
  CYCLE 1 DAY 8 |  |  |  |  | 24.46 (32.10) |  | 31.96 (32.79) |

24. Secondary Outcome: AUC (0-504h) for Belantamab Mafodotin ADC, Treatment B
Description: as for outcome 17
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post Dose on Cycle 1 Day 1; Cycle 1 Day 4; Cycle 1 Day 8; Cycle 1 Day 11; Cycle 1 Day 21
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 7 | 10 | 4 | 7 | 7 | 15 | 8 | 11
h*ug/mL | 6129.71 (23.83) | 4451.74 (23.33) | 6073.99 (37.06) | 5395.98 (20.49) | 4341.73 (22.36) | 5013.84 (31.91) | 5702.03 (26.30) | 6230.16 (35.02)

25. Secondary Outcome: AUC (0-1008h) for Belantamab Mafodotin ADC, Treatment B
Description: Blood samples were collected at indicated timepoints for PK analysis. PK parameter was determined using standard non-compartmental methods. AUC(0-1008h) was derived only for Belantamab mafodotin 1.9 mg/kg STRETCH + Bor/Dex, Belantamab mafodotin 2.5 mg/kg StepDown STRETCH + Bor/Dex and Belantamab mafodotin 2.5 mg/kg STRETCH + Bor/Dex cohorts.
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post Dose on Cycle 1 Day 1; Cycle 1 Day 4; Cycle 1 Day 11; Cycle 1 Day 22; Pre-Dose and Post-Dose on Week 5 Day 7
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points have been analyzed. As per protocol, blood sampling for PK was performed for only specified treatment arms for this OM and hence there are 0 participants analyzed for rest of the arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Groups:
- Belantamab Mafodotin 1.9mg/kg SINGLE+ Bor/Dex: Participants with RRMM received belantamab mafodotin as SINGLE full dose of 1.9mg/kg on Day 1 of every 21-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC/IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles.
- Belantamab Mafodotin 2.5mg/kg SPLIT +Bor/Dex: Participants with RRMM received belantamab mafodotin as two equal divided doses of a total 2.5mg/kg dose as a 1.25mg/kg on Day 1 and 1.25 mg/kg dose on Day 8 of every 21-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC/IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9,11, and 12 of every 21-day cycle up to 8 cycles.
- Belantamab Mafodotin 2.5mg/kg SINGLE+ Bor/Dex: Participants with RRMM received belantamab mafodotin as SINGLE full dose of 2.5mg/kg on Day 1 of every 21-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC/IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles.
- Belantamab Mafodotin 3.4mg/kg SPLIT +Bor/Dex: Participants with RRMM received belantamab mafodotin as two equal divided doses of a total 3.4mg/kg dose as a 1.7 mg/kg dose on Day 1 and 1.7 mg/kg on Day 8 of every 21-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC/IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles.
- Belantamab Mafodotin 3.4mg/kg SINGLE+ Bor/Dex: Participants with RRMM received belantamab mafodotin as SINGLE full dose of 3.4mg/kg on Day 1 of every 21-day cycle as a 30-60 minute infusion. Along with belantamab mafodotin, Bortezomib was administered as 1.3 mg/m^2 SC/IV on Days 1, 4, 8, and 11 with 20 mg Dexamethasone PO/IV on Days 1, 2, 4, 5, 8, 9, 11, and 12 of every 21-day cycle up to 8 cycles.
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Belantamab Mafodotin 1.9mg/kg SINGLE+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Belantamab Mafodotin 2.5mg/kg SPLIT +Bor/Dex | Belantamab Mafodotin 2.5mg/kg SINGLE+ Bor/Dex | Belantamab Mafodotin 3.4mg/kg SPLIT +Bor/Dex | Belantamab Mafodotin 3.4mg/kg SINGLE+ Bor/Dex
Number analyzed (Participants) | 5 | 0 | 10 | 6 | 0 | 0 | 0 | 0
h*ug/mL | 7084.63 (24.82) |  | 7396.49 (25.94) | 6487.41 (26.24) |  |  |  |

26. Secondary Outcome: Tmax for Belantamab Mafodotin ADC, Treatment B
Description: as for outcome 17
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 17
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Hour
  CYCLE 1 DAY 1: number analyzed (Participants) | 12 | 12 | 12 | 12 | 13 | 18 | 11 | 16
  CYCLE 1 DAY 1 | 1.900 [0.63 to 22.50] | 1.125 [0.55 to 2.62] | 2.025 [0.63 to 25.95] | 1.175 [0.62 to 2.57] | 1.233 [0.50 to 2.22] | 1.308 [0.45 to 2.70] | 0.583 [0.50 to 2.20] | 2.000 [0.52 to 3.83]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 0 | 12 | 0
  CYCLE 1 DAY 8 |  |  |  |  | 0.733 [0.52 to 336.75] |  | 0.642 [0.40 to 2.05] |

27. Secondary Outcome: Tlast for Belantamab Mafodotin ADC, Treatment B
Description: as for outcome 20
Time Frame: Pre-Dose Cycle 1 Day 1 to pre-dose Cycle 5 Day 1
Population: as for outcome 17
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Hour | 540.250 [75.67 to 1052.33] | 505.592 [503.75 to 1220.95] | 1009.933 [500.93 to 1489.00] | 755.442 [22.68 to 2018.57] | 504.567 [144.83 to 1351.17] | 506.817 [167.50 to 577.33] | 503.458 [239.72 to 1584.50] | 506.092 [2.00 to 2022.58]

28. Secondary Outcome: Ctrough for Belantamab Mafodotin ADC, Treatment B
Description: as for outcome 17
Time Frame: Pre-Dose, Post-Dose 0, 2 and 24 Hour on Cycle 1 Day 1 and Cycle 1 Day 8; Pre-Dose and Post-Dose on Week 4 Day 1, Week 7 Day 1, Week 10 Day 1, Week 13 Day 1, Week 13 Day 8
Population: as for outcome 17
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 4 | 11 | 4 | 5 | 12 | 15 | 12 | 14
ug/mL
  CYCLE 1 DAY 1 | 1.12 [0.5 to 1.5] | 1.92 [0.6 to 3.9] | 0.63 [0.5 to 1.2] | 0.84 [0.5 to 1.0] | 3.50 [1.8 to 7.1] | 2.12 [1.1 to 5.4] | 4.25 [1.6 to 11.7] | 2.10 [0.5 to 4.3]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 0 | 10 | 0
  CYCLE 1 DAY 8 |  |  |  |  | 3.72 [0.7 to 24.3] |  | 3.93 [1.7 to 9.0] |
  WEEK 4 DAY 1: number analyzed (Participants) | 0 | 8 | 0 | 0 | 5 | 10 | 5 | 5
  WEEK 4 DAY 1 |  | 3.23 [1.4 to 5.4] |  |  | 4.39 [3.0 to 8.6] | 1.32 [0.6 to 8.6] | 3.62 [1.4 to 6.2] | 2.53 [0.6 to 4.3]
  WEEK 7 DAY 1: number analyzed (Participants) | 1 | 5 | 3 | 2 | 4 | 3 | 3 | 0
  WEEK 7 DAY 1 | NA [1.7 to 1.7] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 3.90 [0.5 to 6.4] | 1.24 [0.6 to 2.8] | NA [0.7 to 1.9] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 5.85 [4.0 to 8.1] | 2.72 [0.1 to 3.7] | 10.10 [5.7 to 13.9] |
  WEEK 10 DAY 1: number analyzed (Participants) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1
  WEEK 10 DAY 1 |  |  | NA [0.6 to 0.7] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [6.6 to 6.6] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [4.9 to 4.9] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [4.9 to 4.9] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  WEEK 13 DAY 1: number analyzed (Participants) | 1 | 0 | 3 | 2 | 0 | 1 | 1 | 2
  WEEK 13 DAY 1 | NA [3.2 to 3.2] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | 1.40 [0.7 to 2.1] | NA [2.0 to 3.4] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [6.3 to 6.3] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [10.3 to 10.3] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [1.5 to 5.7] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  WEEK 13 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WEEK 13 DAY 8 |  |  |  |  |  |  | NA [1.7 to 1.7] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |

29. Secondary Outcome: C-EOI for Belantamab Mafodotin ADC, Treatment B
Description: as for outcome 17
Time Frame: Pre-Dose, Post-Dose 0, 2 and 24 Hour on Cycle 1 Day 1 and Cycle 1 Day 8; Pre-Dose and Post-Dose on Week 4 Day 1, Week 7 Day 1, Week 7 Day 8, Week 7 Day 11, Week 10 Day 1, Week 10 Day 8, Week 13 Day 1, Week 13 Day 8
Population: as for outcome 17
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
ug/mL
  CYCLE 1 DAY 1: number analyzed (Participants) | 12 | 12 | 12 | 12 | 13 | 18 | 11 | 16
  CYCLE 1 DAY 1 | 44.75 [26.8 to 68.0] | 44.05 [36.1 to 61.5] | 52.00 [22.8 to 88.8] | 45.25 [31.4 to 76.7] | 22.30 [12.9 to 30.6] | 45.80 [29.1 to 57.6] | 30.10 [11.0 to 49.1] | 54.85 [37.2 to 215.0]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 0 | 12 | 0
  CYCLE 1 DAY 8 |  |  |  |  | 22.60 [12.2 to 48.4] |  | 32.60 [17.5 to 55.7] |
  WEEK 4 DAY 1: number analyzed (Participants) | 0 | 11 | 0 | 0 | 9 | 17 | 9 | 10
  WEEK 4 DAY 1 |  | 46.00 [30.5 to 64.0] |  |  | 27.10 [16.7 to 32.4] | 44.50 [26.8 to 254.0] | 26.20 [14.6 to 53.2] | 51.20 [45.7 to 57.8]
  WEEK 7 DAY 1: number analyzed (Participants) | 5 | 8 | 6 | 7 | 5 | 8 | 5 | 4
  WEEK 7 DAY 1 | 48.60 [37.9 to 83.6] | 44.30 [3.4 to 71.8] | 36.45 [26.5 to 76.9] | 42.50 [25.9 to 84.1] | 26.30 [19.1 to 29.7] | 31.70 [18.2 to 62.7] | 27.40 [12.1 to 38.6] | 38.35 [37.0 to 55.8]
  WEEK 7 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
  WEEK 7 DAY 8 |  |  |  |  | NA [21.0 to 32.6] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [37.0 to 45.1] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |
  WEEK 7 DAY 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WEEK 7 DAY 11 |  |  |  |  |  |  | NA [19.1 to 19.1] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |
  WEEK 10 DAY 1: number analyzed (Participants) | 0 | 0 | 3 | 1 | 2 | 0 | 1 | 1
  WEEK 10 DAY 1 |  |  | 38.00 [31.9 to 43.3] | NA [81.8 to 81.8] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [24.9 to 33.2] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [28.7 to 28.7] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [60.3 to 60.3] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  WEEK 10 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WEEK 10 DAY 8 |  |  |  |  | NA [28.2 to 28.2] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  |  |
  WEEK 13 DAY 1: number analyzed (Participants) | 1 | 1 | 5 | 2 | 0 | 2 | 1 | 3
  WEEK 13 DAY 1 | NA [33.3 to 33.3] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [46.9 to 46.9] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 43.30 [31.1 to 60.1] | NA [70.8 to 95.7] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [33.5 to 43.5] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [27.9 to 27.9] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 46.60 [41.4 to 62.3]
  WEEK 13 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WEEK 13 DAY 8 |  |  |  |  |  |  | NA [37.0 to 37.0] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |

30. Secondary Outcome: Cmax for Belantamab Mafodotin (Total Antibody), Treatment A
Description: as for outcome 17
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16
ug/mL
  CYCLE 1 DAY 1 | 43.09 (22.26) | 40.18 (13.23) | 26.64 (14.97) | 46.95 (30.63)
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 12 | 0
  CYCLE 1 DAY 8 |  |  | 35.11 (13.68) |

31. Secondary Outcome: AUC (0-504h) for Belantamab Mafodotin (Total Antibody), Treatment A
Description: as for outcome 17
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1; Cycle 1 Day 4; Cycle 1 Day 8; Cycle 1 Day 11; Cycle 1 Day 15-21
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 4 | 4 | 10 | 9
h*ug/mL | 6648.19 (35.67) | 6607.45 (35.62) | 6909.91 (24.70) | 7277.25 (28.00)

32. Secondary Outcome: AUC (0-672h) for Belantamab Mafodotin (Total Antibody), Treatment A
Description: as for outcome 17
Time Frame: as for outcome 18
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 4 | 4 | 10 | 9
h*ug/mL | 7408.65 (36.03) | 7249.58 (39.00) | 7828.12 (27.15) | 8146.00 (28.29)

33. Secondary Outcome: AUC (0-1008h) for Belantamab Mafodotin (Total Antibody), Treatment A
Description: Blood samples were collected at indicated timepoints for PK analysis. PK parameter was determined using standard non-compartmental methods. AUC(0-1008) was derived only for Belantamab mafodotin 1.9mg/kg + Len/Dex STRETCH cohort.
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1; Cycle 1 Day 4; Cycle 1 Day 8; Cycle 1 Day 29; Pre-Dose and Post-Dose on Week 5 Day 7
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex
Number analyzed (Participants) | 5
h*ug/mL | 8143.85 (30.12)

34. Secondary Outcome: AUC(0-1344h) for Belantamab Mafodotin (Total Antibody), Treatment A
Description: Blood samples were collected at indicated timepoints for PK analysis. PK parameter was determined using standard non-compartmental methods. AUC(0-1344) was derived only for Belantamab mafodotin 1.9mg/kg + Len/Dex STRETCH cohort.
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1; Cycle 1 Day 4; Cycle 1 Day 8; Cycle 1 Day 29; Pre-Dose and Post-Dose on Week 7 Day 7
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex
Number analyzed (Participants) | 5
h*ug/mL | 8633.05 (30.26)

35. Secondary Outcome: Tmax for Belantamab Mafodotin (Total Antibody), Treatment A
Description: as for outcome 17
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 17
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16
Hour
  CYCLE 1 DAY 1 | 1.267 [0.57 to 2.37] | 1.342 [0.50 to 2.17] | 1.033 [0.57 to 2.20] | 2.000 [0.53 to 2.82]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 12 | 0
  CYCLE 1 DAY 8 |  |  | 1.583 [0.57 to 2.10] |

36. Secondary Outcome: Tlast for Belantamab Mafodotin (Total Antibody), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods. Tlast is the time of last observed quantifiable concentration of belantamab mafodotin in Cycle 1 which extended beyond protocol defined duration for some participants across treatment groups.
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1 and Cycle 1 Day 4; Cycle 1 Day 8; Cycle 1 Day 11; Cycle 1 Day 15-21; Cycle 1 Day 29; pre-dose Cycle 2 Day 28; pre-dose Cycle 3 Day 8
Population: as for outcome 17
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16
Hour | 657.267 [25.50 to 1439.63] | 685.875 [673.92 to 697.75] | 674.833 [670.60 to 1416.93] | 673.625 [2.00 to 1534.15]

37. Secondary Outcome: Ctrough for Belantamab Mafodotin (Total Antibody), Treatment A
Description: as for outcome 17
Time Frame: Pre-Dose, Post-Dose 0, 2 and 24 Hour on Cycle 1 Day 1 and Cycle 1 Day 8; Pre-Dose and Post-Dose on Week 5 Day 1, Week 5 Day 8, Week 9 Day 1, Week 9 Day 8, Week 13 Day 1, Week 13 Day 8
Population: as for outcome 17
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 4 | 4 | 12 | 12
ug/mL
  CYCLE 1 DAY 1 | 0.81 [0.6 to 2.0] | 3.39 [0.7 to 6.1] | 7.74 [1.9 to 9.9] | 3.16 [1.6 to 5.9]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 11 | 0
  CYCLE 1 DAY 8 |  |  | 3.99 [0.9 to 12.3] |
  WEEK 5 DAY 1: number analyzed (Participants) | 0 | 3 | 9 | 5
  WEEK 5 DAY 1 |  | 2.76 [1.1 to 8.1] | 12.40 [7.7 to 22.6] | 1.82 [0.8 to 4.5]
  WEEK 5 DAY 8: number analyzed (Participants) | 0 | 0 | 7 | 0
  WEEK 5 DAY 8 |  |  | 6.16 [2.5 to 22.6] |
  WEEK 9 DAY 1: number analyzed (Participants) | 1 | 1 | 6 | 2
  WEEK 9 DAY 1 | NA [2.7 to 2.7] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [8.7 to 8.7] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 15.25 [11.2 to 29.7] | NA [10.4 to 11.0] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  WEEK 9 DAY 8: number analyzed (Participants) | 0 | 0 | 3 | 0
  WEEK 9 DAY 8 |  |  | 10.50 [1.3 to 10.5] |
  WEEK 13 DAY 1: number analyzed (Participants) | 2 | 0 | 2 | 3
  WEEK 13 DAY 1 | NA [1.6 to 2.4] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [12.1 to 19.2] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 10.70 [0.9 to 17.0]
  WEEK 13 DAY 8: number analyzed (Participants) | 0 | 0 | 1 | 0
  WEEK 13 DAY 8 |  |  | NA [10.5 to 10.5] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |

38. Secondary Outcome: C-EOI for Belantamab Mafodotin (Total Antibody), Treatment A
Description: as for outcome 17
Time Frame: as for outcome 37
Population: as for outcome 17
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 10 | 4 | 12 | 16
ug/mL
  CYCLE 1 DAY 1: number analyzed (Participants) | 10 | 3 | 12 | 16
  CYCLE 1 DAY 1 | 42.70 [35.0 to 64.0] | 36.90 [35.3 to 47.9] | 27.25 [20.1 to 32.7] | 47.00 [17.2 to 64.2]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 12 | 0
  CYCLE 1 DAY 8 |  |  | 35.00 [27.8 to 40.3] |
  WEEK 5 DAY 1: number analyzed (Participants) | 0 | 4 | 9 | 10
  WEEK 5 DAY 1 |  | 42.15 [32.4 to 48.1] | 27.00 [24.7 to 36.4] | 45.70 [30.0 to 79.9]
  WEEK 5 DAY 8: number analyzed (Participants) | 0 | 0 | 9 | 0
  WEEK 5 DAY 8 |  |  | 36.40 [27.8 to 50.6] |
  WEEK 9 DAY 1: number analyzed (Participants) | 6 | 1 | 8 | 2
  WEEK 9 DAY 1 | 41.80 [33.1 to 52.9] | NA [44.4 to 44.4] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 31.25 [22.9 to 46.6] | NA [38.6 to 52.1] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  WEEK 9 DAY 8: number analyzed (Participants) | 0 | 0 | 6 | 0
  WEEK 9 DAY 8 |  |  | 39.20 [27.4 to 56.8] |
  WEEK 13 DAY 1: number analyzed (Participants) | 1 | 0 | 2 | 4
  WEEK 13 DAY 1 | NA [28.1 to 28.1] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [24.0 to 36.3] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 50.10 [39.5 to 73.3]
  WEEK 13 DAY 8: number analyzed (Participants) | 0 | 0 | 2 | 0
  WEEK 13 DAY 8 |  |  | NA [32.3 to 44.8] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |

39. Secondary Outcome: Cmax for Belantamab Mafodotin (Total Antibody) Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 10 | 12 | 12 | 13 | 17 | 11 | 16
ug/mL
  CYCLE 1 DAY 1: number analyzed (Participants) | 12 | 10 | 12 | 12 | 13 | 17 | 10 | 16
  CYCLE 1 DAY 1 | 41.28 (16.86) | 37.47 (12.02) | 53.29 (23.50) | 53.85 (12.54) | 22.92 (35.83) | 50.32 (30.03) | 31.06 (20.02) | 78.29 (36.16)
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 11 | 0 | 11 | 0
  CYCLE 1 DAY 8 |  |  |  |  | 29.47 (40.48) |  | 45.31 (39.57) |

40. Secondary Outcome: AUC (0-504h) for Belantamab Mafodotin (Total Antibody), Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post Dose on Cycle 1 Day 1; Cycle 1 Day 4; Cycle 1 Day 8; Cycle 1 Day 11; Cycle 1 Day 21
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 8 | 6 | 4 | 6 | 8 | 12 | 7 | 11
h*ug/mL | 7310.17 (37.27) | 6094.55 (33.37) | 8386.87 (25.44) | 9891.43 (29.93) | 8283.76 (32.51) | 8207.69 (41.72) | 9812.19 (27.13) | 12581.08 (28.13)

41. Secondary Outcome: AUC (0-1008h) for Belantamab Mafodotin (Total Antibody), Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods. AUC(0-1008h) was derived only for Belantamab mafodotin 1.9 mg/kg STRETCH + Bor/Dex, Belantamab mafodotin 2.5 mg/kg StepDown STRETCH + Bor/Dex and Belantamab mafodotin 2.5 mg/kg STRETCH + Bor/Dex cohorts.
Time Frame: as for outcome 25
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex
Number analyzed (Participants) | 5 | 11 | 10
h*ug/mL | 11656.56 (25.11) | 11328.37 (40.25) | 11178.97 (49.10)

42. Secondary Outcome: Tmax for Belantamab Mafodotin (Total Antibody), Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 17
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 10 | 12 | 12 | 13 | 17 | 11 | 16
Hour
  CYCLE 1 DAY 1: number analyzed (Participants) | 12 | 10 | 12 | 12 | 13 | 17 | 10 | 16
  CYCLE 1 DAY 1 | 1.900 [0.75 to 2.03] | 2.033 [0.70 to 2.23] | 0.983 [0.57 to 2.13] | 1.142 [0.62 to 2.58] | 2.000 [0.50 to 2.17] | 1.983 [0.45 to 2.23] | 0.650 [0.50 to 2.13] | 2.000 [0.52 to 2.50]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 11 | 0 | 11 | 0
  CYCLE 1 DAY 8 |  |  |  |  | 0.700 [0.52 to 2.50] |  | 0.617 [0.40 to 2.05] |

43. Secondary Outcome: Tlast for Belantamab Mafodotin (Total Antibody), Treatment B
Description: as for outcome 36
Time Frame: Pre-Dose Cycle 1 Day 1 to pre-dose Cycle 9 Day 1
Population: as for outcome 17
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Hour | 585.958 [75.67 to 2855.48] | 504.983 [239.92 to 2155.95] | 1414.500 [505.25 to 3694.62] | 1031.467 [1006.72 to 4054.38] | 504.583 [144.83 to 1351.17] | 505.483 [167.50 to 671.65] | 502.883 [239.72 to 717.68] | 506.808 [2.00 to 2832.25]

44. Secondary Outcome: Ctrough for Belantamab Mafodotin (Total Antibody), Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, Post-Dose 0, 2 and 24 Hour on Cycle 1 Day 1 and Cycle 1 Day 8; Pre-Dose and Post-Dose on Week 4 Day 1, Week 7 Day 1, Week 7 Day 8, Week 10 Day 1, Week 13 Day 1, Week 13 Day 8
Population: as for outcome 17
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 4 | 10 | 9 | 11 | 12 | 14 | 12 | 15
ug/mL
  CYCLE 1 DAY 1: number analyzed (Participants) | 4 | 9 | 9 | 11 | 12 | 14 | 12 | 15
  CYCLE 1 DAY 1 | 3.13 [1.0 to 5.6] | 5.27 [2.1 to 10.7] | 1.53 [1.1 to 4.5] | 1.32 [0.6 to 8.6] | 5.88 [1.2 to 13.5] | 7.22 [1.7 to 17.2] | 9.59 [3.5 to 38.9] | 6.82 [1.4 to 17.4]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 0 | 8 | 0
  CYCLE 1 DAY 8 |  |  |  |  | 12.30 [2.7 to 33.2] |  | 12.05 [7.8 to 22.6] |
  WEEK 4 DAY 1: number analyzed (Participants) | 0 | 10 | 0 | 0 | 6 | 12 | 5 | 8
  WEEK 4 DAY 1 |  | 7.97 [0.6 to 18.8] |  |  | 14.95 [1.2 to 27.7] | 3.62 [0.6 to 22.8] | 11.20 [5.3 to 25.1] | 5.27 [1.9 to 13.2]
  WEEK 7 DAY 1: number analyzed (Participants) | 2 | 6 | 5 | 3 | 4 | 5 | 3 | 0
  WEEK 7 DAY 1 | NA [2.7 to 5.7] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 7.66 [2.6 to 22.2] | 1.72 [1.4 to 6.5] | 2.32 [1.9 to 5.8] | 19.40 [10.3 to 34.0] | 1.35 [1.1 to 21.7] | 26.00 [19.1 to 31.0] |
  WEEK 7 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WEEK 7 DAY 8 |  |  |  |  | NA [1.5 to 1.5] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  |  |
  WEEK 10 DAY 1: number analyzed (Participants) | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 1
  WEEK 10 DAY 1 |  |  | 3.07 [1.4 to 3.4] | NA [2.3 to 2.3] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [16.6 to 16.6] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [20.7 to 20.7] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [23.0 to 23.0] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  WEEK 13 DAY 1: number analyzed (Participants) | 1 | 0 | 4 | 2 | 0 | 1 | 1 | 2
  WEEK 13 DAY 1 | NA [12.0 to 12.0] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | 5.26 [1.3 to 10.5] | NA [9.3 to 14.5] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [32.3 to 32.3] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [29.2 to 29.2] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [10.0 to 18.9] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  WEEK 13 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WEEK 13 DAY 8 |  |  |  |  |  |  | NA [10.0 to 10.0] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |

45. Secondary Outcome: C-EOI for Belantamab Mafodotin (Total Antibody), Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, Post-Dose 0, 2 and 24 Hour on Cycle 1 Day 1 and Cycle 1 Day 8; Pre-Dose and Post-Dose on Week 4 Day 1, Week 7 Day 1, Week 7 Day 8, Week 7 Day 11, Week 10 Day 1, Week 13 Day 1, Week 13 Day 8
Population: as for outcome 17
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 11 | 11 | 12 | 12 | 12 | 16 | 11 | 15
ug/mL
  CYCLE 1 DAY 1: number analyzed (Participants) | 11 | 10 | 12 | 12 | 12 | 14 | 9 | 15
  CYCLE 1 DAY 1 | 36.60 [30.7 to 52.0] | 36.75 [27.6 to 44.0] | 52.55 [38.2 to 90.3] | 51.65 [43.7 to 66.1] | 23.90 [13.9 to 33.1] | 44.35 [30.3 to 63.0] | 33.40 [21.2 to 40.1] | 68.80 [42.5 to 241.0]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0 | 11 | 0
  CYCLE 1 DAY 8 |  |  |  |  | 24.95 [16.1 to 38.2] |  | 42.50 [25.7 to 98.9] |
  WEEK 4 DAY 1: number analyzed (Participants) | 0 | 11 | 0 | 0 | 8 | 16 | 7 | 10
  WEEK 4 DAY 1 |  | 39.20 [24.6 to 54.6] |  |  | 37.00 [19.8 to 46.0] | 59.50 [30.1 to 233.0] | 39.40 [19.6 to 70.8] | 67.85 [50.0 to 85.5]
  WEEK 7 DAY 1: number analyzed (Participants) | 5 | 8 | 6 | 8 | 5 | 8 | 5 | 4
  WEEK 7 DAY 1 | 36.50 [31.8 to 67.8] | 43.00 [14.3 to 78.6] | 37.30 [23.3 to 65.1] | 47.50 [33.3 to 67.7] | 42.00 [24.0 to 49.5] | 50.75 [29.6 to 73.8] | 33.90 [20.2 to 63.0] | 63.95 [44.5 to 67.6]
  WEEK 7 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
  WEEK 7 DAY 8 |  |  |  |  | NA [32.2 to 60.4] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [46.5 to 82.0] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |
  WEEK 7 DAY 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WEEK 7 DAY 11 |  |  |  |  |  |  | NA [34.9 to 34.9] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |
  WEEK 10 DAY 1: number analyzed (Participants) | 0 | 0 | 3 | 1 | 2 | 0 | 1 | 1
  WEEK 10 DAY 1 |  |  | 42.70 [41.0 to 53.6] | NA [64.6 to 64.6] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [31.6 to 44.2] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [36.9 to 36.9] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [61.1 to 61.1] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  WEEK 10 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WEEK 10 DAY 8 |  |  |  |  | NA [40.7 to 40.7] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  |  |
  WEEK 13 DAY 1: number analyzed (Participants) | 1 | 1 | 5 | 2 | 0 | 2 | 1 | 3
  WEEK 13 DAY 1 | NA [37.0 to 37.0] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [29.6 to 29.6] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 33.30 [27.8 to 41.6] | NA [68.4 to 72.8] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [37.6 to 51.2] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [49.5 to 49.5] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 54.50 [52.9 to 85.3]
  WEEK 13 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WEEK 13 DAY 8 |  |  |  |  |  |  | NA [48.0 to 48.0] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |

46. Secondary Outcome: Cmax for Belantamab Mafodotin Cysteine Maleimidocaproyl Monomethyl Auristatin F (Cys-mcMMAF), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 11 | 4 | 12 | 13
ug/mL
  CYCLE 1 DAY 1 | 1.11 (70.59) | 0.55 (53.90) | 0.53 (48.23) | 1.18 (53.35)
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 12 | 0
  CYCLE 1 DAY 8 |  |  | 0.63 (28.28) |

47. Secondary Outcome: AUC (0-168h) for Belantamab Mafodotin (Cys-mcMMAF), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose, 0, 2, and 24 Hours Post Dose on Cycle 1 Day 1, and Cycle 1 Day 8
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 9 | 1 | 11 | 10
h*ug/mL
  CYCLE 1 DAY 1 | 106.21 (55.99) | NA (NA) — As pre-specified in the SAP, data is not reported if the number of participants analyzed is less than 3. | 43.15 (26.42) | 113.58 (49.61)
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 8 | 0
  CYCLE 1 DAY 8 |  |  | 51.31 (30.45) |

48. Secondary Outcome: AUC (0-336h) for Belantamab Mafodotin (Cys-mcMMAF), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods. AUC (0-336h) was derived only for the Belantamab mafodotin 2.5mg/kg + Len/Dex SPLIT cohort.
Time Frame: Pre-dose, 0, 2, and 24 Hours Post Dose on Cycle 1 Day 1; Cycle 1 Day 4; Cycle 1 Day 8; Cycle 1 Day 11; Cycle 1 Day 14
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex
Number analyzed (Participants) | 8
h*ug/mL | 93.84 (29.16)

49. Secondary Outcome: Tmax for Belantamab Mafodotin (Cys-mcMMAF), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 17
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 11 | 4 | 12 | 13
Hour
  CYCLE 1 DAY 1 | 24.217 [1.42 to 28.58] | 24.900 [23.67 to 73.42] | 23.667 [1.00 to 25.42] | 24.367 [2.23 to 25.92]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 12 | 0
  CYCLE 1 DAY 8 |  |  | 23.425 [0.57 to 25.93] |

50. Secondary Outcome: Tlast for Belantamab Mafodotin (Cys-mcMMAF), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose Cycle 1 Day 1 to pre-dose Cycle 1 Day 15
Population: as for outcome 17
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 14
Hour | 165.567 [25.50 to 357.02] | 120.283 [49.97 to 191.58] | 336.900 [94.40 to 360.17] | 166.167 [2.08 to 239.17]

51. Secondary Outcome: C-EOI for Belantamab Mafodotin (Cys-mcMMAF), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, Post-Dose 0, 2 and 24 Hour on Cycle 1 Day 1 and Cycle 1 Day 8; Pre-Dose and Post-Dose on Week 5 Day 1, Week 7 Day 8, Week 9 Day 1, Week 9 Day 8, Week 13 Day 1, Week 13 Day 8
Population: as for outcome 17
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 11 | 4 | 13 | 14
ug/mL
  CYCLE 1 DAY 1 | 0.43 [0.3 to 1.6] | 0.187 [0.160 to 0.290] | 0.19 [0.1 to 1.3] | 0.29 [0.1 to 1.3]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 12 | 0
  CYCLE 1 DAY 8 |  |  | 0.29 [0.2 to 0.9] |
  WEEK 5 DAY 1: number analyzed (Participants) | 0 | 4 | 8 | 10
  WEEK 5 DAY 1 |  | 0.16 [0.1 to 0.4] | 0.13 [0.1 to 0.3] | 0.28 [0.2 to 1.0]
  WEEK 7 DAY 8: number analyzed (Participants) | 0 | 0 | 7 | 0
  WEEK 7 DAY 8 |  |  | 0.23 [0.2 to 0.4] |
  WEEK 9 DAY 1: number analyzed (Participants) | 6 | 1 | 8 | 2
  WEEK 9 DAY 1 | 0.29 [0.2 to 0.5] | NA [0.1 to 0.1] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 0.13 [0.1 to 0.7] | NA [0.2 to 0.2] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  WEEK 9 DAY 8: number analyzed (Participants) | 0 | 0 | 6 | 0
  WEEK 9 DAY 8 |  |  | 0.24 [0.2 to 0.4] |
  WEEK 13 DAY 1: number analyzed (Participants) | 1 | 0 | 2 | 4
  WEEK 13 DAY 1 | NA [0.4 to 0.4] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [0.1 to 0.2] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 0.68 [0.2 to 0.9]
  WEEK 13 DAY 8: number analyzed (Participants) | 0 | 0 | 3 | 0
  WEEK 13 DAY 8 |  |  | 0.243 [0.207 to 0.248] |

52. Secondary Outcome: Cmax for Belantamab Mafodotin (Cys-mcMMAF) Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 10 | 12 | 12 | 12 | 11 | 11 | 11 | 9
ug/mL
  CYCLE 1 DAY 1 | 0.73 (29.88) | 0.75 (68.94) | 1.03 (52.77) | 1.29 (38.95) | 0.65 (87.99) | 1.15 (57.18) | 1.03 (38.56) | 1.09 (40.30)
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 0 | 10 | 0
  CYCLE 1 DAY 8 |  |  |  |  | 0.58 (87.48) |  | 0.86 (64.55) |

53. Secondary Outcome: AUC(0-168h) for Belantamab Mafodotin (Cys-mcMMAF), Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose, 0, 2, and 24 Hours Post Dose on Cycle 1 Day 1, Cycle 1 Day 4; and Cycle 1 Day 7
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 0 | 0 | 8 | 0 | 9 | 0 | 10 | 0
h*ug/mL |  |  | 89.05 (41.52) |  | 52.82 (96.74) |  | 81.17 (31.46) |

54. Secondary Outcome: Tmax for Belantamab Mafodotin (Cys-mcMMAF), Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0, 2 and 24 Hours Post-Dose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 17
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 10 | 12 | 12 | 12 | 11 | 11 | 11 | 9
Hour
  CYCLE 1 DAY 1 | 22.225 [22.07 to 24.77] | 24.475 [1.00 to 25.75] | 23.092 [22.00 to 25.95] | 22.442 [1.17 to 74.02] | 24.083 [19.30 to 77.37] | 24.083 [2.07 to 25.25] | 24.583 [22.97 to 70.28] | 24.667 [21.85 to 25.72]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 0 | 10 | 0
  CYCLE 1 DAY 8 |  |  |  |  | 24.000 [0.92 to 25.30] |  | 23.717 [2.58 to 25.60] |

55. Secondary Outcome: Tlast for Belantamab Mafodotin (Cys-mcMMAF), Treatment B
Description: as for outcome 36
Time Frame: Pre-Dose Cycle 1 Day 1 to pre-dose Cycle 2 Day 1
Population: as for outcome 17
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Hour | 85.542 [68.57 to 262.25] | 239.800 [72.33 to 243.90] | 237.992 [70.58 to 265.82] | 93.942 [67.95 to 242.77] | 241.283 [146.33 to 527.50] | 237.425 [70.53 to 241.58] | 240.675 [237.55 to 503.73] | 171.567 [2.00 to 266.87]

56. Secondary Outcome: C-EOI for Belantamab Mafodotin (Cys-mcMMAF), Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: as for outcome 29
Population: as for outcome 17
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 13 | 17 | 11 | 15
ug/mL
  CYCLE 1 DAY 1 | 0.29 [0.1 to 0.5] | 0.21 [0.1 to 2.7] | 0.28 [0.2 to 0.6] | 0.32 [0.1 to 1.4] | 0.19 [0.1 to 0.7] | 0.29 [0.1 to 0.8] | 0.27 [0.1 to 0.8] | 0.39 [0.2 to 0.6]
  CYCLE 1 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 12 | 0 | 11 | 0
  CYCLE 1 DAY 8 |  |  |  |  | 0.27 [0.1 to 1.5] |  | 0.40 [0.2 to 0.9] |
  WEEK 4 DAY 1: number analyzed (Participants) | 0 | 10 | 0 | 0 | 9 | 16 | 9 | 10
  WEEK 4 DAY 1 |  | 0.19 [0.1 to 0.4] |  |  | 0.21 [0.1 to 0.4] | 0.35 [0.1 to 1.5] | 0.26 [0.2 to 0.6] | 0.35 [0.2 to 0.9]
  WEEK 7 DAY 1: number analyzed (Participants) | 6 | 7 | 6 | 8 | 5 | 7 | 5 | 4
  WEEK 7 DAY 1 | 0.20 [0.1 to 0.4] | 0.21 [0.1 to 0.3] | 0.17 [0.1 to 0.2] | 0.31 [0.1 to 0.9] | 0.27 [0.1 to 0.4] | 0.24 [0.1 to 0.9] | 0.20 [0.2 to 0.4] | 0.36 [0.2 to 0.4]
  WEEK 7 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
  WEEK 7 DAY 8 |  |  |  |  | NA [0.2 to 0.3] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [0.3 to 0.6] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |
  WEEK 7 DAY 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WEEK 7 DAY 11 |  |  |  |  |  |  | NA [5.0 to 5.0] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |
  WEEK 10 DAY 1: number analyzed (Participants) | 0 | 0 | 3 | 1 | 2 | 0 | 1 | 1
  WEEK 10 DAY 1 |  |  | 0.236 [0.188 to 0.238] | NA [0.5 to 0.5] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [0.2 to 0.4] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [0.3 to 0.3] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [0.4 to 0.4] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  WEEK 10 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WEEK 10 DAY 8 |  |  |  |  | NA [1.6 to 1.6] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  |  |
  WEEK 13 DAY 1: number analyzed (Participants) | 2 | 0 | 5 | 2 | 0 | 2 | 1 | 3
  WEEK 13 DAY 1 | NA [0.1 to 0.4] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | 0.222 [0.118 to 0.240] | NA [0.4 to 0.4] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [0.2 to 0.6] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | NA [0.3 to 0.3] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 0.24 [0.1 to 0.3]
  WEEK 13 DAY 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WEEK 13 DAY 8 |  |  |  |  |  |  | NA [0.3 to 0.3] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |

57. Secondary Outcome: Cmax for Lenalidomide (25 mg), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0.5, 1, 2, 4 and 24 hours on Cycle 1 Day 1 post lenalidomide dose
Population: Pharmacokinetic (PK) population. Only those participants who received 25 mg lenalidomide with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 5 | 4 | 0 | 13
ug/mL | 382.16 (54.52) | 331.53 (17.91) |  | 283.08 (36.55)

58. Secondary Outcome: AUC(0-24h) for Lenalidomide (25 mg), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0.5, 1, 2, 4 and 24 hours on Cycle 1 Day 1 post lenalidomide dose
Population: as for outcome 57
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 4 | 3 | 0 | 8
h*ug/mL | 2247.36 (65.76) | 1577.62 (21.66) |  | 2117.26 (38.21)

59. Secondary Outcome: AUC (0-4h) for Lenalidomide (25 mg), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0.5, 1, 2 and 4 hours on Cycle 1 Day 1 post lenalidomide dose
Population: as for outcome 57
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 5 | 3 | 0 | 9
h*ug/mL | 812.22 (105.88) | 870.92 (19.36) |  | 620.10 (44.84)

60. Secondary Outcome: Tmax for Lenalidomide (25 mg), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0.5, 1, 2, 4 and 24 hours on Cycle 1 Day 1 post lenalidomide dose
Population: as for outcome 57
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 5 | 4 | 0 | 13
Hour | 0.967 [0.47 to 4.00] | 1.417 [0.93 to 2.00] |  | 3.767 [1.92 to 4.00]

61. Secondary Outcome: Tlast for Lenalidomide (25 mg), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, Post dose on Cycle 1 Day 1
Population: as for outcome 57
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 5 | 4 | 0 | 13
Hour | 20.750 [3.80 to 24.00] | 4.000 [3.77 to 22.57] |  | 22.050 [3.75 to 23.55]

62. Secondary Outcome: Cmax for Lenalidomide (10 mg), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0.5, 1, 2, 4 and 24 hours on Cycle 1 Day 1 post lenalidomide dose
Population: Pharmacokinetic (PK) population. Only those participants who received 10 mg lenalidomide with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 4 | 0 | 0 | 2
ug/mL | 193.06 (36.86) |  |  | NA (NA) — As pre-specified in the SAP, data is not reported if the number of participants analyzed is less than 3.

63. Secondary Outcome: AUC(0-24h) for Lenalidomide (10 mg), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0.5, 1, 2, 4 and 24 hours on Cycle 1 Day 1 post lenalidomide dose
Population: as for outcome 62
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 4 | 0 | 0 | 1
h*ug/mL | 1660.82 (22.40) |  |  | NA (NA) — As pre-specified in the SAP, data is not reported if the number of participants analyzed is less than 3.

64. Secondary Outcome: AUC (0-4h) for Lenalidomide (10 mg), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0.5, 1, 2 and 4 hours on Cycle 1 Day 1 post lenalidomide dose
Population: as for outcome 62
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 4 | 0 | 0 | 2
h*ug/mL | 486.46 (41.84) |  |  | NA (NA) — As pre-specified in the SAP, data is not reported if the number of participants analyzed is less than 3.

65. Secondary Outcome: Tmax for Lenalidomide (10 mg), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0.5, 1, 2, 4 and 24 hours on Cycle 1 Day 1 post lenalidomide dose
Population: as for outcome 62
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 4 | 0 | 0 | 2
Hour | 2.000 [0.53 to 3.80] |  |  | NA [1.13 to 4.00] — As pre-specified in the SAP, data is not reported if the number of participants analyzed is less than 3.

66. Secondary Outcome: Tlast for Lenalidomide (10 mg), Treatment A
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, Post dose on Cycle 1 Day 1
Population: as for outcome 62
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex
Number analyzed (Participants) | 4 | 0 | 0 | 2
Hour | 21.583 [21.27 to 23.68] |  |  | NA [4.00 to 4.00] — As pre-specified in the SAP, data is not reported if the number of participants analyzed is less than 3.

67. Secondary Outcome: Cmax for Bortezomib, Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, 0.5, 1, 2, 4 and 24 Hours Post-Dose on Cycle 1 Day 1
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points for Bortezomib have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 0 | 11 | 0 | 0 | 0 | 15 | 0 | 15
ug/mL
  INTRAVENOUS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  INTRAVENOUS |  |  |  |  |  | NA (NA) — As pre-specified in the SAP, data is not reported if the number of participants analyzed is less than 3. |  | NA (NA) — As pre-specified in the SAP, data is not reported if the number of participants analyzed is less than 3.
  SUBCUTANEOUS |  | 14.45 (50.16) |  |  |  | 14.89 (44.03) |  | 15.88 (42.07)

68. Secondary Outcome: AUC (0-72h) for Bortezomib, Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose, 5 minute, 0.25, 0.5, 1, 2, 4, 6, 10, 24, 48 and 72 hour post bortezomib dose
Population: Pharmacokinetic (PK) population. Only those participants who received Bortezomib with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 0 | 11 | 0 | 0 | 0 | 14 | 0 | 13
h*ug/mL
  Intravenous: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Intravenous |  |  |  |  |  | NA (NA) — As pre-specified in the SAP, data is not reported if the number of participants analyzed is less than 3. |  | NA (NA) — As pre-specified in the SAP, data is not reported if the number of participants analyzed is less than 3.
  Subcutaneous |  | 95.10 (21.71) |  |  |  | 73.03 (30.79) |  | 73.06 (21.57)

69. Secondary Outcome: AUC (0-t) for Bortezomib, Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose, 5 minute, 0.25, 0.5, 1, 2, 4, 6, 10, 24, 48 and 72 hour post bortezomib dose
Population: as for outcome 68
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 0 | 11 | 0 | 0 | 0 | 15 | 0 | 15
h*ug/mL
  Intravenous: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Intravenous |  |  |  |  |  | NA (NA) — As pre-specified in the SAP, data is not reported if the number of participants analyzed is less than 3. |  | NA (NA) — As pre-specified in the SAP, data is not reported if the number of participants analyzed is less than 3.
  Subcutaneous |  | 89.48 (25.50) |  |  |  | 69.51 (31.87) |  | 71.70 (26.79)

70. Secondary Outcome: Tmax for Bortezomib, Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose, 5 minute, 0.25, 0.5, 1, 2, 4, 6, 10, 24, 48 and 72 hour post bortezomib dose
Population: as for outcome 68
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 0 | 11 | 0 | 0 | 0 | 15 | 0 | 15
Hour
  Intravenous: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Intravenous |  |  |  |  |  | NA [0.08 to 0.08] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [0.13 to 0.13] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  Subcutaneous |  | 0.533 [0.10 to 1.07] |  |  |  | 0.517 [0.25 to 1.00] |  | 0.500 [0.08 to 1.00]

71. Secondary Outcome: Tlast for Bortezomib, Treatment B
Description: Blood samples were collected for PK analysis. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-Dose, Post dose on Cycle 1 Day 3
Population: as for outcome 68
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 0 | 11 | 0 | 0 | 1 | 16 | 0 | 15
Hour
  Intravenous: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Intravenous |  |  |  |  |  | NA [46.97 to 46.97] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. |  | NA [70.52 to 70.52] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3.
  Subcutaneous |  | 68.867 [44.07 to 72.00] |  |  | NA [73.07 to 73.07] — As pre-specified in the SAP, median is not reported if the number of participants analyzed is less than 3. | 68.392 [44.35 to 73.10] |  | 48.000 [46.17 to 75.65]

72. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADAs) Against Belantamab Mafodotin
Description: Serum samples were collected and tested for the presence of antibodies against belantamab mafodotin using validated immunoassays.
Time Frame: Up to approximately 4.5 years (End of Treatment [EoT])
Population: All Treated. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 3 | 13 | 15 | 12 | 12 | 12 | 12 | 12 | 18 | 11 | 16
Participants
  Baseline (Day 1) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  EoT (Up to approx. 4.5 years): number analyzed (Participants) | 3 | 3 | 8 | 5 | 4 | 6 | 4 | 10 | 5 | 11 | 7 | 11
  EoT (Up to approx. 4.5 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

73. Secondary Outcome: Titers of ADAs Against Belantamab Mafodotin
Description: Serum samples were collected and tested for the presence of antibodies against belantamab mafodotin using validated immunoassays. Confirmed positive ADA samples were further analyzed to obtain the titer of the antibodies. Titers of anti-drug antibodies against belantamab mafodotin is presented.
Time Frame: Up to approximately 4.5 years
Population: All Treated. Only those participants with data available at specified time points have been analyzed. There were no participants with positive ADA results at end of treatment. Hence the titer (concentration) of ADA was not collected.
Measure: Median (Full Range); unit: Titers
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Titers |  |  |  | 100 [NA to NA] — Full range is not applicable as only a single participant was analyzed. Median value presented here is the actual titer value for this single participant. |  |  |  |  | 100 [NA to NA] — Full range is not applicable as only a single participant was analyzed. Median value presented here is the actual titer value for this single participant. |  | 100 [NA to NA] — Full range is not applicable as only a single participant was analyzed. Median value presented here is the actual titer value for this single participant. |

74. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI) Total Scores
Description: The OSDI is a 12-item questionnaire designed to assess both the frequency of dry eye symptoms and their impact on vision-related functioning. OSDI consist of three subscales (ocular symptoms: item 1-3; visual related function: item 4-9; environmental triggers: item 10-12). Each item will be graded on a scale of 0 (none of the time or lower disability) to 4 (all of the time or greater disability) with total scores ranging from 0 (no disability) to 100 (complete disability). The total OSDI score was calculated as (sum of scores for all questions answered*100) divided by (total number of questions answered*4). Higher scores indicated greater disability. Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All Treated. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 9 | 4 | 11 | 12 | 12 | 9 | 12 | 9 | 10 | 15 | 9 | 14
Score on scale
  Baseline (Day 1) | 11.1 (7.58) | 0.8 (1.56) | 7.8 (9.30) | 11.4 (14.26) | 10.8 (17.20) | 2.4 (2.79) | 7.8 (9.94) | 8.0 (5.66) | 12.4 (16.42) | 6.3 (7.71) | 8.6 (13.61) | 3.3 (5.58)
  Change from baseline (up to approx. 4.5 years): number analyzed (Participants) | 2 | 3 | 4 | 5 | 5 | 4 | 6 | 7 | 2 | 9 | 5 | 7
  Change from baseline (up to approx. 4.5 years) | -5.2 (4.42) | 0.6 (4.10) | 6.9 (12.03) | 2.2 (7.19) | 15.2 (35.94) | 15.9 (14.80) | 18.7 (34.95) | 29.3 (39.18) | 6.1 (8.59) | 14.4 (23.26) | 48.3 (27.42) | 19.3 (14.41)

75. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) Overall Composite Scores
Description: The NEI-VFQ-25 consisted of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question to assess the patient's perception of vision-related functioning and vision-related quality of life. Items were coded to a 0 to 100 scale and were averaged to calculate domains. The composite score ranges from 0 (worst score) to 100 (best score), with higher scores indicating better vision-related functioning. Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All Treated. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 10 | 3 | 11 | 12 | 11 | 8 | 9 | 8 | 7 | 11 | 7 | 10
Score on scale
  Baseline (Day 1) | 85.1 (11.42) | 89.0 (18.43) | 91.9 (10.88) | 91.0 (11.35) | 88.0 (16.92) | 95.5 (4.70) | 96.2 (5.20) | 95.3 (4.60) | 90.4 (7.67) | 94.1 (8.33) | 93.2 (7.13) | 94.7 (5.59)
  Change from baseline (up to approx. 4.5 years): number analyzed (Participants) | 3 | 2 | 4 | 5 | 4 | 4 | 4 | 6 | 1 | 6 | 3 | 5
  Change from baseline (up to approx. 4.5 years) | 0.2 (13.53) | 12.9 (22.42) | -4.5 (4.04) | -1.9 (3.43) | 1.1 (19.48) | -8.4 (13.65) | -18.3 (19.96) | -26.0 (31.54) | 1.3 | -13.2 (25.00) | -48.9 (2.35) | -11.5 (15.39)

76. Secondary Outcome: Number of Participants With Symptomatic AEs Measured by Patient-reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: The PRO-CTCAE is a patient-reported outcome measure developed to evaluate symptomatic toxicity in participants on cancer clinical trials. It included item library of 124 items representing 78 symptomatic toxicities drawn from the CTCAE like Anxious, Blurred Vision, Chills, Concentration, Constipation, Cough, Decreased Appetite, Discouraged, Dizziness, Fatigue, Heart Palpitations, Insomnia, Memory, Mouth/Throat Sores, Nausea, Nosebleed, Numbness & Tingling, Pain, Ringing In Ears, Shortness Of Breath, Vomiting and Watery Eyes. Number of participants with symptomatic AEs measured by PRO-CTCAEs are presented.
Time Frame: Up to approximately 4.5 years
Population: All Treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Participants
  Anxious | 8 | 4 | 13 | 13 | 8 | 12 | 12 | 11 | 11 | 17 | 10 | 15
  Blurred Vision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills | 8 | 4 | 13 | 13 | 8 | 12 | 12 | 11 | 11 | 17 | 10 | 15
  Concentration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Constipation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cough | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Decreased Appetite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Discouraged | 8 | 4 | 13 | 13 | 8 | 12 | 12 | 11 | 11 | 17 | 10 | 15
  Dizziness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Heart Palpitations | 8 | 4 | 13 | 13 | 8 | 12 | 12 | 11 | 11 | 17 | 10 | 15
  Insomnia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Memory | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mouth/Throat Sores | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea | 8 | 4 | 13 | 13 | 8 | 12 | 12 | 11 | 11 | 17 | 10 | 15
  Nosebleed | 8 | 4 | 13 | 13 | 8 | 12 | 12 | 11 | 11 | 17 | 10 | 15
  Numbness & tingling | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain | 8 | 4 | 13 | 13 | 8 | 12 | 12 | 11 | 11 | 17 | 10 | 15
  Ringing In Ears | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Shortness Of Breath | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vomiting | 8 | 4 | 13 | 13 | 8 | 12 | 12 | 11 | 11 | 17 | 10 | 15
  Watery Eyes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

77. Secondary Outcome: Number of Participants With AEs of Special Interest (AESI)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Number of participants with AESI for belantamab mafodotin (corneal events, thrombocytopenia and infusion related reactions) are presented.
Time Frame: Up to approximately 4.5 years
Population: All Treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Participants
  AESI (Corneal Events) | 9 | 3 | 12 | 11 | 9 | 12 | 12 | 12 | 10 | 17 | 10 | 16
  AESI (Thrombocytopenia) | 4 | 2 | 7 | 11 | 9 | 12 | 10 | 11 | 11 | 13 | 12 | 14
  AESI (Infusion Related Reactions) | 1 | 0 | 2 | 3 | 0 | 2 | 1 | 2 | 2 | 3 | 3 | 1

78. Secondary Outcome: Number of Participants With Worst-case Change From Baseline in Best Corrected Visual Acuity Test (BCVA) Scores
Description: BCVA score was assessed individually for each eye. BCVA score was calculated based on the Logarithm of the Minimum Angle of Resolution (logMAR score). Any worst-case change from baseline categories are presented for right and left eyes. BCVA test scores were categorized as no change/improved vision, possible worsened vision and definite worsened vision. No change/improved vision was defined as a change from baseline <0.12 logMAR score; a possible worsened vision was defined as a change from baseline >=0.12 to <0.3 logMAR score; a definite worsened vision was defined as a change from baseline >=0.3 logMAR score. Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All Treated. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 9 | 4 | 13 | 14 | 11 | 12 | 12 | 12 | 12 | 18 | 11 | 16
Participants
  Right Eye, No change/improved vision | 2 | 2 | 5 | 3 | 4 | 3 | 2 | 2 | 4 | 3 | 2 | 1
  Right Eye, Possible worsened vision | 3 | 0 | 0 | 2 | 2 | 2 | 0 | 4 | 2 | 2 | 5 | 5
  Right Eye, Definite worsened vision | 4 | 2 | 8 | 9 | 5 | 7 | 10 | 6 | 6 | 13 | 4 | 10
  Left Eye, No change/improved vision | 2 | 1 | 2 | 4 | 4 | 1 | 2 | 5 | 4 | 3 | 3 | 2
  Left Eye, Possible worsened vision | 2 | 0 | 2 | 1 | 0 | 3 | 5 | 1 | 2 | 3 | 2 | 6
  Left Eye, Definite worsened vision | 5 | 3 | 9 | 9 | 7 | 8 | 5 | 6 | 6 | 12 | 6 | 8

79. Secondary Outcome: Number of Participants With Worst-case Post-baseline Change in BCVA Scores by Snellen Results
Description: BCVA score was assessed individually for better seeing eye and worse seeing eye. BCVA score was calculated based on the Logarithm of the Minimum Angle of Resolution (logMAR score). Any worst-case change post baseline categories are presented for better seeing eye and worse seeing eye. BCVA test scores by Snellen results were categorized as improved BCVA, <= 2 lines decline in visual acuity from baseline, >= 3 lines decline in visual acuity from baseline. Number of lines change from baseline was defined as the following: Improved BCVA equates to a negative change in logMAR from baseline BCVA. <= 2 lines decline in visual acuity equates to logMAR change from baseline ≤0.37. >= 3 lines decline in visual acuity equates to logMAR change from baseline ≥0.38. Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All Treated. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 9 | 4 | 13 | 14 | 11 | 12 | 12 | 12 | 12 | 18 | 11 | 16
Participants
  Better seeing Eye, Improved BCVA | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Better seeing Eye, <=2 Lines decline in visual acuity from baseline | 8 | 3 | 9 | 11 | 7 | 7 | 10 | 8 | 9 | 8 | 9 | 12
  Better seeing Eye, >=3 Lines decline in visual acuity from baseline | 1 | 1 | 3 | 3 | 4 | 5 | 2 | 4 | 2 | 9 | 2 | 4
  Worse seeing Eye, Improved BCVA | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Worse seeing Eye, <=2 Lines decline in visual acuity from baseline | 5 | 3 | 4 | 5 | 6 | 5 | 8 | 7 | 6 | 6 | 7 | 8
  Worse seeing Eye, >=3 Lines decline in visual acuity from baseline | 4 | 1 | 8 | 9 | 4 | 7 | 4 | 5 | 5 | 12 | 4 | 8

80. Secondary Outcome: Number of Participants With Post-baseline Decline in BCVA to Light Perception or no Light Perception
Description: Number of participants with a Decline in BCVA to 'Light Perception (LP)' or 'No Light Perception (NLP)' due to a Corneal Event Anytime Post-Baseline are presented. BCVA score was assessed individually for each eye (Left and Right). Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits. Number of participants analyzed were who have any post-baseline BCVA score, where the Visual Acuity is due to corneal findings.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All Treated. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 9 | 3 | 10 | 11 | 11 | 10 | 12 | 11 | 8 | 11 | 8 | 10
Participants
  Left Eye, LP: number analyzed (Participants) | 8 | 3 | 10 | 11 | 9 | 10 | 12 | 11 | 8 | 11 | 7 | 9
  Left Eye, LP | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Left Eye, NLP: number analyzed (Participants) | 8 | 3 | 10 | 11 | 9 | 10 | 12 | 11 | 8 | 11 | 7 | 9
  Left Eye, NLP | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Right Eye, LP | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Right Eye, NLP | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

81. Secondary Outcome: Number of Participants With Shift in Corneal Epithelium Findings From no (Baseline) to Yes (Worst Post-Baseline)
Description: Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits. Corneal epithelium findings like active edema, active opacity, corneal neovascularization (CN), corneal ulcer, epithelial microcystic edema (EME) and subepithelial haze were performed using a slit lamp. Number of participants with shift in corneal epithelium findings from no (Baseline) to yes (worst post-Baseline) are presented.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All Treated. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 12 | 4 | 13 | 16 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 16
Participants
  Active Edema, Right Eye | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Active Edema, Left Eye | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Active Opacity, Right Eye: number analyzed (Participants) | 12 | 3 | 13 | 16 | 12 | 12 | 12 | 12 | 12 | 18 | 12 | 16
  Active Opacity, Right Eye | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
  Active Opacity, Left Eye: number analyzed (Participants) | 12 | 4 | 12 | 16 | 12 | 12 | 12 | 12 | 13 | 18 | 12 | 15
  Active Opacity, Left Eye | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
  Corneal Neovascularization, Right Eye: number analyzed (Participants) | 12 | 4 | 13 | 16 | 11 | 12 | 11 | 12 | 13 | 17 | 12 | 16
  Corneal Neovascularization, Right Eye | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Corneal Neovascularization, Left Eye: number analyzed (Participants) | 12 | 4 | 13 | 16 | 11 | 12 | 12 | 11 | 12 | 17 | 12 | 16
  Corneal Neovascularization, Left Eye | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Corneal Ulcer, Right Eye: number analyzed (Participants) | 12 | 3 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 14 | 12 | 16
  Corneal Ulcer, Right Eye | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Corneal Ulcer, Left Eye: number analyzed (Participants) | 12 | 3 | 13 | 14 | 12 | 12 | 12 | 12 | 13 | 14 | 12 | 16
  Corneal Ulcer, Left Eye | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Epithelial Microcystic Edema, Right Eye | 2 | 1 | 3 | 6 | 2 | 3 | 3 | 3 | 3 | 9 | 3 | 9
  Epithelial Microcystic Edema, Left Eye | 2 | 2 | 2 | 6 | 4 | 3 | 4 | 2 | 4 | 8 | 3 | 9
  Subepithelial Haze, Right Eye: number analyzed (Participants) | 11 | 3 | 13 | 16 | 12 | 12 | 12 | 12 | 12 | 18 | 12 | 16
  Subepithelial Haze, Right Eye | 3 | 1 | 5 | 8 | 5 | 8 | 3 | 6 | 5 | 9 | 8 | 9
  Subepithelial Haze, Left Eye: number analyzed (Participants) | 11 | 4 | 13 | 16 | 12 | 12 | 12 | 12 | 12 | 18 | 12 | 16
  Subepithelial Haze, Left Eye | 3 | 2 | 6 | 9 | 6 | 9 | 5 | 4 | 4 | 10 | 8 | 10

82. Secondary Outcome: Number of Participants With Worse Grade Post-baseline Punctate Keratopathy Findings
Description: Participants with worse grade punctate keratopathy findings post baseline at any ocular exam by right eye, left eye and worse eye are presented as none, mild, moderate and severe. Worse eye indicates the eye with the worst visual acuity. Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years
Population: All Treated. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 9 | 4 | 13 | 14 | 11 | 12 | 12 | 12 | 12 | 18 | 11 | 16
Participants
  Right Eye, None | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1
  Right Eye, Mild | 1 | 2 | 5 | 6 | 5 | 3 | 5 | 1 | 2 | 3 | 2 | 2
  Right Eye, Moderate | 5 | 2 | 3 | 6 | 5 | 7 | 4 | 7 | 5 | 9 | 6 | 9
  Right Eye, Severe | 1 | 0 | 3 | 2 | 1 | 1 | 3 | 4 | 3 | 6 | 2 | 4
  Left Eye, None | 1 | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 2 | 0 | 1 | 0
  Left Eye, Mild | 3 | 2 | 1 | 4 | 5 | 3 | 5 | 2 | 1 | 3 | 2 | 2
  Left Eye, Moderate | 4 | 2 | 9 | 6 | 3 | 5 | 5 | 5 | 7 | 9 | 6 | 10
  Left Eye, Severe | 1 | 0 | 1 | 4 | 1 | 2 | 2 | 5 | 2 | 6 | 2 | 4
  Worst eye, None | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0
  Worst eye, Mild | 1 | 2 | 1 | 4 | 5 | 3 | 5 | 1 | 1 | 2 | 2 | 2
  Worst eye, Moderate | 6 | 2 | 7 | 6 | 5 | 6 | 3 | 6 | 6 | 10 | 6 | 9
  Worst eye, Severe | 1 | 0 | 3 | 4 | 1 | 2 | 4 | 5 | 3 | 6 | 2 | 5

83. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30-item Core Module (EORTC QLQ-C30) Score
Description: The EORTC QLQ-C30 includes 30-items with single and multi-item scales. These included five functional scales (physical functioning [PF], role functioning [RF], cognitive functioning [CF], emotional functioning [EF] and social functioning [SF]), three symptom scales (fatigue, pain and nausea/vomiting [N/V]), a global health status (GHS)/ Quality-of-Life (QoL) scale, and six single items (constipation, diarrhea, insomnia, dyspnea, appetite loss [AL] and financial difficulties [FD]). Response options are 1 to 4. Scores were averaged and transformed to 0 to 100, a high score for functional scales/ GHS/QoL represent better functioning ability or health-related quality-of-life (HRQoL), whereas a high score for symptom scales/ single items represent significant symptomatology. Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits. Change from Baseline (CFB) was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years (End of treatment [EoT])
Population: All Treated. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 10 | 3 | 10 | 8 | 12 | 9 | 11 | 11 | 9 | 10 | 10 | 8
Score on scale
  GHS/QoL, Baseline (Day 1) | 65.8 (25.29) | 69.4 (31.55) | 58.3 (14.16) | 60.4 (13.18) | 56.2 (23.33) | 67.6 (9.72) | 63.6 (20.84) | 56.1 (20.78) | 60.2 (26.61) | 55.0 (24.60) | 63.3 (16.29) | 67.7 (15.71)
  GHS/QoL, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  GHS/QoL, CFB to EoT | -50.0 (22.05) | 4.2 (17.68) | -4.2 (14.43) | -16.7 (18.00) | -10.0 (34.05) | -8.3 (11.79) | 0.0 (13.94) | -14.6 (25.88) | -4.2 (17.68) | -8.3 (9.62) | 18.7 (23.94) | 4.2 (20.97)
  PF, Baseline (Day 1) | 67.3 (23.82) | 88.9 (13.88) | 78.7 (15.65) | 73.3 (21.97) | 75.0 (15.60) | 84.4 (17.95) | 85.5 (17.34) | 70.9 (25.69) | 66.7 (31.27) | 78.7 (19.58) | 82.0 (10.91) | 89.4 (11.48)
  PF, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  PF, CFB to EoT | -17.8 (48.23) | 13.3 (18.86) | -6.7 (24.94) | 0.0 (33.11) | -5.3 (22.80) | -10.0 (14.14) | -1.1 (9.81) | -12.5 (27.93) | 3.3 (4.71) | -10.0 (15.87) | -11.7 (42.64) | -1.7 (12.62)
  RF, Baseline (Day 1) | 66.7 (30.43) | 88.9 (19.25) | 76.7 (22.50) | 72.9 (29.46) | 68.1 (21.86) | 72.2 (22.05) | 81.8 (24.10) | 57.6 (36.03) | 70.4 (33.10) | 73.3 (19.56) | 71.7 (22.29) | 89.6 (19.80)
  RF, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  RF, CFB to EoT | -22.2 (69.39) | 16.7 (23.57) | 8.3 (34.69) | 4.2 (34.36) | -6.7 (25.28) | -8.3 (35.36) | -11.1 (27.22) | 0.0 (32.12) | 0.0 (0.00) | -20.8 (34.36) | 20.8 (36.96) | -4.2 (28.46)
  EF, Baseline (Day 1) | 76.7 (25.40) | 86.1 (4.81) | 77.5 (18.02) | 76.0 (16.93) | 70.8 (20.87) | 94.4 (7.22) | 73.5 (25.50) | 68.9 (28.89) | 83.3 (13.18) | 78.3 (17.21) | 83.3 (16.20) | 91.7 (8.91)
  EF, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  EF, CFB to EoT | 5.6 (29.27) | -12.5 (5.89) | 0.0 (0.00) | 10.4 (15.77) | 3.3 (33.64) | -16.7 (23.57) | 0.0 (11.79) | -6.3 (25.49) | -12.5 (5.89) | 2.1 (14.23) | -12.5 (15.96) | 6.3 (12.50)
  CF, Baseline (Day 1) | 75.0 (16.20) | 88.9 (9.62) | 71.7 (24.91) | 72.9 (21.71) | 81.9 (19.41) | 87.0 (13.89) | 81.8 (17.41) | 74.2 (15.57) | 74.1 (16.90) | 83.3 (22.22) | 95.0 (8.05) | 91.7 (12.60)
  CF, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  CF, CFB to EoT | -16.7 (44.10) | 8.3 (11.79) | 16.7 (19.25) | 12.5 (20.97) | -10.0 (25.28) | -16.7 (23.57) | 2.8 (6.80) | 0.0 (17.82) | 8.3 (11.79) | -8.3 (21.52) | -16.7 (27.22) | -8.3 (9.62)
  SF, Baseline (Day 1) | 71.7 (26.12) | 88.9 (19.25) | 80.0 (18.92) | 77.1 (21.71) | 76.4 (20.67) | 83.3 (18.63) | 77.3 (28.16) | 71.2 (28.95) | 72.2 (34.36) | 68.3 (34.65) | 73.3 (17.92) | 75.0 (23.57)
  SF, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  SF, CFB to EoT | -27.8 (63.10) | 8.3 (11.79) | 0.0 (23.57) | -12.5 (36.96) | -6.7 (25.28) | -16.7 (0.00) | -11.1 (22.77) | -27.1 (36.66) | 0.0 (0.00) | 8.3 (16.67) | -12.5 (34.36) | 16.7 (19.25)
  Fatigue, Baseline (Day 1) | 46.7 (23.89) | 25.9 (16.97) | 31.1 (8.76) | 38.9 (19.70) | 34.3 (19.22) | 28.4 (21.60) | 29.3 (13.40) | 34.3 (26.51) | 30.9 (30.32) | 32.2 (23.10) | 37.8 (25.77) | 31.9 (3.93)
  Fatigue, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  Fatigue, CFB to EoT | 3.7 (35.72) | -11.1 (15.71) | 5.6 (6.42) | 2.8 (24.64) | 13.3 (28.76) | -11.1 (15.71) | -3.7 (13.46) | 16.7 (33.60) | 11.1 (15.71) | 2.8 (18.98) | -2.8 (41.94) | -11.1 (12.83)
  N/V, Baseline (Day 1) | 11.7 (15.81) | 0.0 (0.00) | 11.7 (15.81) | 2.1 (5.89) | 8.3 (15.08) | 3.7 (7.35) | 4.5 (7.78) | 1.5 (5.03) | 5.6 (8.33) | 8.3 (11.79) | 5.0 (8.05) | 2.1 (5.89)
  N/V, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  N/V, CFB to EoT | 11.1 (41.94) | 0.0 (0.00) | 4.2 (8.33) | -4.2 (8.33) | -6.7 (30.28) | -8.3 (11.79) | 5.6 (17.21) | 6.3 (12.40) | 0.0 (0.00) | -4.2 (8.33) | 4.2 (8.33) | 0.0 (13.61)
  Pain, Baseline (Day 1) | 46.7 (35.83) | 22.2 (25.46) | 36.7 (24.60) | 37.5 (31.81) | 41.7 (26.11) | 24.1 (29.00) | 28.8 (25.92) | 34.8 (34.52) | 42.6 (33.45) | 28.3 (20.86) | 36.7 (25.82) | 22.9 (21.71)
  Pain, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  Pain, CFB to EoT | 0.0 (16.67) | -16.7 (47.14) | -12.5 (15.96) | -25.0 (50.00) | 20.0 (36.13) | -16.7 (23.57) | -5.6 (8.61) | 12.5 (30.54) | -8.3 (11.79) | 25.0 (31.91) | -4.2 (43.83) | 8.3 (16.67)
  Dyspnoea, Baseline (Day 1) | 33.3 (35.14) | 11.1 (19.25) | 13.3 (17.21) | 12.5 (17.25) | 22.2 (25.95) | 11.1 (16.67) | 15.2 (17.41) | 33.3 (36.51) | 14.8 (24.22) | 16.7 (17.57) | 16.7 (17.57) | 8.3 (15.43)
  Dyspnoea, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  Dyspnoea, CFB to EoT | 33.3 (33.33) | -16.7 (23.57) | 25.0 (31.91) | 16.7 (19.25) | 0.0 (23.57) | 0.0 (0.00) | -5.6 (13.61) | 12.5 (39.59) | 16.7 (23.57) | 0.0 (0.00) | 16.7 (19.25) | 0.0 (0.00)
  Insomnia, Baseline (Day 1) | 40.0 (26.29) | 44.4 (38.49) | 33.3 (27.22) | 29.2 (21.36) | 36.1 (33.21) | 25.9 (14.70) | 27.3 (25.03) | 33.3 (33.33) | 37.0 (38.89) | 33.3 (31.43) | 30.0 (33.15) | 8.3 (15.43)
  Insomnia, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  Insomnia, CFB to EoT | 0.0 (33.33) | 0.0 (47.14) | -16.7 (19.25) | 0.0 (27.22) | -6.7 (27.89) | -16.7 (23.57) | 5.6 (25.09) | 8.3 (23.57) | 0.0 (47.14) | -16.7 (19.25) | 0.0 (54.43) | 0.0 (0.00)
  AL, Baseline (Day 1) | 23.3 (27.44) | 0.0 (0.00) | 6.7 (14.05) | 25.0 (23.57) | 13.9 (22.29) | 7.4 (14.70) | 12.1 (16.82) | 9.1 (15.57) | 22.2 (23.57) | 26.7 (26.29) | 6.7 (14.05) | 12.5 (24.80)
  AL, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  AL, CFB to EoT | 22.2 (19.25) | 16.7 (23.57) | 16.7 (19.25) | -16.7 (19.25) | 0.0 (33.33) | 16.7 (23.57) | 0.0 (0.00) | -4.2 (21.36) | 0.0 (0.00) | -8.3 (41.94) | 25.0 (50.00) | -8.3 (16.67)
  Constipation, Baseline (Day 1) | 20.0 (28.11) | 0.0 (0.00) | 6.7 (14.05) | 12.5 (17.25) | 16.7 (26.59) | 11.1 (16.67) | 12.1 (16.82) | 9.1 (15.57) | 7.4 (22.22) | 13.3 (17.21) | 20.0 (32.20) | 8.3 (15.43)
  Constipation, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  Constipation, CFB to EoT | 0.0 (0.00) | 16.7 (23.57) | 16.7 (33.33) | 16.7 (33.33) | 0.0 (0.00) | 0.0 (47.14) | 0.0 (0.00) | 4.2 (21.36) | 0.0 (0.00) | 0.0 (0.00) | -25.0 (31.91) | 16.7 (19.25)
  Diarrhoea, Baseline (Day 1) | 6.7 (14.05) | 0.0 (0.00) | 16.7 (23.57) | 8.3 (15.43) | 19.4 (22.29) | 11.1 (16.67) | 9.1 (15.57) | 21.2 (34.23) | 11.1 (33.33) | 6.7 (21.08) | 6.7 (14.05) | 12.5 (17.25)
  Diarrhoea, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  Diarrhoea, CFB to EoT | 22.2 (19.25) | 33.3 (47.14) | 8.3 (31.91) | 8.3 (16.67) | -13.3 (29.81) | -16.7 (23.57) | -5.6 (13.61) | 0.0 (30.86) | 0.0 (0.00) | 0.0 (27.22) | 16.7 (19.25) | -8.3 (31.91)
  FD, Baseline (Day 1) | 30.0 (33.15) | 11.1 (19.25) | 30.0 (36.68) | 0.0 (0.00) | 36.1 (30.01) | 7.4 (14.70) | 24.2 (36.79) | 15.2 (17.41) | 25.9 (27.78) | 26.7 (37.84) | 20.0 (35.83) | 20.8 (35.36)
  FD, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 8 | 2 | 4 | 4 | 4
  FD, CFB to EoT | 33.3 (57.74) | 0.0 (0.00) | 8.3 (31.91) | 0.0 (0.00) | -13.3 (18.26) | 0.0 (0.00) | 0.0 (0.00) | 4.2 (21.36) | 0.0 (0.00) | 16.7 (19.25) | 8.3 (16.67) | -16.7 (33.33)

84. Secondary Outcome: Change From Baseline in EORTC QLQ 20-item Multiple Myeloma Module (MY20) Score
Description: The EORTC QLQ-MY20 is a supplement to the QLQ-C30 instrument used in participants with multiple myeloma. The module comprised of 20 questions that addressed four myeloma-specific HRQoL domains: disease symptoms (DS), side effects of treatment (SET), future perspective (FP) and body image (BI). Responses are 1 to 4. Scores were averaged and scales were transformed to 0 to 100 scale. A high score for disease symptoms and side effects of treatment represented a high level of symptomatology or problems, whereas a high score for future perspective and body image represented better outcomes. Baseline (Day 1) was defined as latest pre-dose assessment with non-missing value, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and up to approximately 4.5 years (End of treatment [EoT])
Population: All Treated. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex
Number analyzed (Participants) | 10 | 3 | 10 | 9 | 12 | 9 | 11 | 9 | 9 | 10 | 10 | 8
Score on scale
  DS, Baseline (Day 1) | 45.0 (25.45) | 24.1 (22.45) | 26.6 (12.22) | 24.7 (19.47) | 40.7 (19.58) | 21.0 (19.40) | 21.2 (17.88) | 31.5 (21.15) | 29.0 (23.37) | 26.7 (15.89) | 25.6 (20.15) | 18.8 (8.88)
  DS, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 7 | 2 | 4 | 4 | 4
  DS, CFB to EoT | -14.8 (17.86) | -8.3 (27.50) | 10.0 (9.34) | -5.6 (36.00) | 23.3 (26.76) | -2.8 (19.64) | -8.3 (10.39) | 5.6 (22.22) | 5.6 (15.71) | -2.8 (18.43) | 12.5 (20.48) | 4.2 (13.13)
  SET, Baseline (Day 1) | 27.5 (16.65) | 21.0 (18.64) | 19.9 (11.20) | 18.8 (13.87) | 23.6 (13.79) | 7.7 (6.87) | 12.7 (9.65) | 15.1 (9.43) | 14.9 (6.21) | 16.7 (14.21) | 13.9 (13.60) | 11.3 (8.99)
  SET, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 7 | 2 | 4 | 4 | 4
  SET, CFB to EoT | -11.4 (15.19) | -14.8 (15.71) | 0.1 (7.86) | 0.0 (9.07) | 0.0 (14.60) | 1.9 (7.86) | 3.3 (5.00) | 19.0 (19.38) | 1.1 (6.81) | -2.7 (8.74) | 5.6 (8.74) | 6.5 (20.14)
  BI, Baseline (Day 1) | 83.3 (17.57) | 100.0 (0.00) | 76.7 (31.62) | 81.5 (24.22) | 77.8 (29.59) | 85.2 (24.22) | 69.7 (37.87) | 88.9 (16.67) | 77.8 (33.33) | 90.0 (22.50) | 93.3 (14.05) | 75.0 (34.50)
  BI, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 7 | 2 | 4 | 4 | 4
  BI, CFB to EoT | -11.1 (50.92) | -16.7 (23.57) | -8.3 (31.91) | 8.3 (41.94) | 6.7 (14.91) | 0.0 (0.00) | 0.0 (0.00) | -9.5 (16.27) | 0.0 (0.00) | -8.3 (16.67) | -8.3 (16.67) | 16.7 (19.25)
  FP, Baseline (Day 1) | 58.9 (29.65) | 48.1 (12.83) | 58.9 (28.71) | 72.8 (16.77) | 65.7 (17.38) | 67.9 (17.07) | 55.6 (31.03) | 59.3 (23.57) | 58.0 (34.15) | 62.2 (15.00) | 63.3 (16.60) | 66.7 (13.28)
  FP, CFB to EoT: number analyzed (Participants) | 3 | 2 | 4 | 4 | 5 | 2 | 6 | 7 | 2 | 4 | 4 | 4
  FP, CFB to EoT | -7.4 (51.32) | 38.9 (39.28) | 16.7 (19.25) | 13.9 (13.98) | -6.7 (21.66) | 0.0 (15.71) | 1.9 (14.77) | -3.2 (22.87) | -5.6 (7.86) | -8.3 (31.91) | -2.8 (44.79) | 22.2 (15.71)

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (non-SAEs) and serious adverse events (SAEs) were collected from Day 1 to Month 53 for Main Study Phase and from Month 53 up to Month 65, which marks the completion of the PACT Phase for all participants.
Description: All treated population included all participants who received at least one dose of study treatment.
Arm/Group | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex | PACT Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex | PACT Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex | PACT Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex | PACT Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex | PACT Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex | PACT Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex | PACT Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex | PACT Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex | PACT Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex | PACT Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex
All-Cause Mortality (participants affected / at risk) | 3/12 | 2/4 | 6/13 | 8/16 | 4/12 | 2/12 | 4/12 | 5/12 | 5/13 | 8/18 | 6/12 | 4/16 | 0/3 | 0/1 | 0/2 | 0/4 | 0/2 | 0/4 | 0/4 | 0/2 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 6/12 | 2/4 | 6/13 | 10/16 | 8/12 | 8/12 | 6/12 | 6/12 | 7/13 | 13/18 | 6/12 | 9/16 | 1/3 | 0/1 | 0/2 | 2/4 | 1/2 | 1/4 | 1/4 | 0/2 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 12/12 | 4/4 | 13/13 | 16/16 | 12/12 | 12/12 | 12/12 | 12/12 | 13/13 | 18/18 | 12/12 | 16/16 | 0/3 | 0/1 | 0/2 | 0/4 | 0/2 | 0/4 | 0/4 | 0/2 | 0/2 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex (N=12) | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex (N=4) | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex (N=13) | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex (N=16) | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex (N=12) | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex (N=12) | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex (N=12) | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex (N=12) | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex (N=13) | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex (N=18) | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex (N=12) | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex (N=16) | PACT Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex (N=3) | PACT Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex (N=1) | PACT Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex (N=2) | PACT Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex (N=4) | PACT Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex (N=2) | PACT Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex (N=4) | PACT Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex (N=4) | PACT Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex (N=2) | PACT Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex (N=2) | PACT Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex (N=1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (5) | 3 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Campylobacter colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic Vein Occlusion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodular regenerative hyperplasia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex (N=12) | Main Study Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex (N=4) | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex (N=13) | Main Study Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex (N=16) | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex (N=12) | Main Study Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex (N=12) | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex (N=12) | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg STRETCH + Bor/Dex (N=12) | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex (N=13) | Main Study Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex (N=18) | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex (N=12) | Main Study Phase: Belantamab Mafodotin 3.4 mg/kg SINGLE + Bor/Dex (N=16) | PACT Phase: Belantamab Mafodotin 1.9mg/kg STRETCH + Len/Dex (N=3) | PACT Phase: Belantamab Mafodotin 1.9mg/kg SINGLE + Len/Dex (N=1) | PACT Phase: Belantamab Mafodotin 2.5mg/kg SPLIT + Len/Dex (N=2) | PACT Phase: Belantamab Mafodotin 2.5mg/kg SINGLE + Len/Dex (N=4) | PACT Phase: Belantamab Mafodotin 1.9 mg/kg STRETCH + Bor/Dex (N=2) | PACT Phase: Belantamab Mafodotin 1.9 mg/kg SINGLE + Bor/Dex (N=4) | PACT Phase: Belantamab Mafodotin 2.5 mg/kg Step-Down STRETCH+ Bor/Dex (N=4) | PACT Phase: Belantamab Mafodotin 2.5 mg/kg SPLIT + Bor/Dex (N=2) | PACT Phase: Belantamab Mafodotin 2.5 mg/kg SINGLE + Bor/Dex (N=2) | PACT Phase: Belantamab Mafodotin 3.4 mg/kg SPLIT + Bor/Dex (N=1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 4 (5) | 5 (5) | 1 (1) | 3 (6) | 2 (2) | 3 (3) | 3 (3) | 4 (5) | 2 (2) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 3 (18) | 2 (3) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 2 (3) | 2 (10) | 2 (2) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (8) | 7 (7) | 4 (8) | 5 (6) | 3 (10) | 5 (9) | 9 (13) | 6 (18) | 9 (10) | 9 (12) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muir-Torre syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (3) | 2 (8) | 1 (2) | 2 (6) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blindness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blindness unilateral (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 (2) | 0 (0) | 1 (1) | 3 (5) | 2 (4) | 2 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract cortical (Eye disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract nuclear (Eye disorders) | 2 (8) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract subcapsular (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (3) | 0 (0) | 2 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cornea verticillata (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal epithelium defect (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal opacity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 (4) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 3 (5) | 1 (2) | 4 (9) | 0 (0) | 4 (7) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (6) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 3 (4) | 4 (10) | 1 (2) | 2 (4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 2 (3) | 0 (0) | 2 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratopathy (Eye disorders) | 9 (114) | 3 (52) | 12 (122) | 11 (224) | 9 (61) | 11 (111) | 12 (123) | 12 (85) | 10 (97) | 15 (188) | 10 (130) | 15 (143) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meibomian gland dysfunction (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (5) | 0 (0) | 2 (6) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night blindness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 4 (9) | 6 (12) | 1 (2) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Posterior capsule opacification (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pterygium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0
Punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 (0) | 1 (2) | 7 (12) | 6 (27) | 1 (2) | 3 (7) | 5 (10) | 5 (9) | 5 (17) | 12 (56) | 3 (6) | 7 (24) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA
Visual acuity reduced (Eye disorders) | 5 (26) | 1 (23) | 4 (29) | 5 (77) | 4 (26) | 6 (39) | 4 (49) | 4 (24) | 1 (2) | 2 (2) | 2 (39) | 3 (7) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 2 (5) | 0 (0) | 2 (3) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aerophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 (3) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 8 (8) | 5 (7) | 2 (2) | 2 (4) | 6 (6) | 0 (0) | 7 (8) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 (9) | 3 (6) | 6 (9) | 6 (11) | 6 (13) | 5 (6) | 6 (11) | 0 (0) | 4 (6) | 8 (12) | 1 (1) | 4 (9) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Loose tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (5) | 3 (4) | 4 (4) | 2 (2) | 5 (5) | 1 (1) | 3 (5) | 8 (18) | 2 (2) | 7 (10) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 2 (2) | 2 (2) | 1 (2) | 2 (2) | 1 (1) | 2 (4) | 3 (4) | 0 (0) | 5 (5) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crepitations (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 (0) | 0 (0) | 4 (5) | 7 (10) | 3 (3) | 5 (6) | 4 (5) | 5 (5) | 4 (5) | 6 (6) | 5 (5) | 3 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (6) | 0 (0) | 2 (2) | 4 (5) | 5 (5) | 2 (2) | 3 (5) | 0 (0) | 5 (5) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Campylobacter colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes ophthalmic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 1 (2) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | 0
Nosocomial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Picornavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (4) | 3 (4) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 9 (11) | 3 (4) | 6 (6) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 (8) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chemical burns of eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 4 (5) | 1 (1) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 | 0 | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 4 (6) | 1 (1) | 3 (5) | 2 (2) | 3 (5) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 1 (2) | 2 (2) | 2 (2) | 3 (7) | 5 (5) | 4 (6) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 2 (2) | 1 (1) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Grip strength decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipids increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 4 (5) | 1 (2) | 4 (9) | 5 (14) | 2 (17) | 2 (2) | 2 (4) | 2 (2) | 1 (2) | 2 (5) | 0 (0) | 1 (4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 3 (3) | 1 (1) | 5 (7) | 4 (6) | 6 (13) | 9 (12) | 7 (12) | 7 (12) | 1 (1) | 9 (11) | 3 (3) | 5 (7) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine albumin/creatinine ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity tests abnormal (Investigations) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (25) | 0 (0) | 3 (13) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appetite disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 1 (1) | 2 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 4 (6) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Magnesium deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (5) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 4 (5) | 3 (3) | 1 (1) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 2 (3) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 5 (5) | 0 (0) | 3 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diffuse idiopathic skeletal hyperostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exposed bone in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (4) | 4 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 4 (6) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (4) | 1 (2) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 3 (3) | 2 (2) | 1 (2) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 3 (5) | 3 (5) | 6 (8) | 3 (5) | 8 (10) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 4 (4) | 1 (2) | 2 (2) | 1 (1) | 4 (6) | 2 (3) | 4 (5) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 5 (6) | 2 (4) | 1 (2) | 6 (7) | 2 (2) | 6 (6) | 3 (3) | 4 (4) | 3 (3) | 6 (6) | 1 (1) | 4 (4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital lesion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2) | 1 (1) | 2 (3) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 4 (4) | 3 (4) | 2 (2) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 4 (5) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 2 (3) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cold urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism venous (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 4 (5) | 2 (2) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT03544281/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT03544281/SAP_001.pdf